

## **Clinical Study Protocol**

DRUG SUBSTANCE(S) VLA1553

VERSION NO. Final 3.0

STUDY CODE VLA1553-302

DATE 07-Apr-2021

A RANDOMIZED, DOUBLE-BLINDED PHASE 3 STUDY TO DEMONSTRATE LOT-TO-LOT CONSISTENCY OF THREE LOTS OF A LIVE-ATTENUATED CHIKUNGUNYA VIRUS VACCINE CANDIDATE (VLA1553) IN HEALTHY ADULTS AGED 18 TO 45 YEARS

Lot-to-Lot study

PROTOCOL NUMBER: VLA1553-302

IND NUMBER: 17854

Sponsor Valneva Austria GmbH

Campus Vienna Biocenter 3 A-1030 Vienna, Austria

NOTE: The information contained in this document is the intelligence property of Valneva Austria GmbH. The privileged and confidential information is intended only for the use of the individual or entity to whom it has been sent or to whom it has been given by a member of Valneva's staff. If the reader of this document is not the intended recipient, you are hereby notified that any dissemination, distribution or copying of this item is strictly prohibited. If you have received this item in error, please notify us by telephone, and immediately return the original and all enclosures to us at Valneva Austria GmbH, Campus Vienna Biocenter 3, 1030 Vienna, Austria.

Valneva Austria GmbH CONFIDENTIAL page 1 / 90

| 1 | PRO" | TOCOL | SIGNA | TURF | PAGE |
|---|------|-------|-------|------|------|

Title of Clinical Trial:

A RANDOMIZED, DOUBLE-BLINDED PHASE 3 STUDY TO DEMONSTRATE LOT-TO-LOT CONSISTENCY OF THREE LOTS OF A LIVE-ATTENUATED CHIKUNGUNYA VIRUS VACCINE CANDIDATE (VLA1553) IN HEALTHY ADULTS AGED 18 TO 45

**YEARS** 

**Protocol Number:** 

VLA1553-302

**IND Number:** 

17854

With their signature, Investigators and Sponsor agree to conduct this study in accordance with the Protocol, International Conference on Harmonization (ICH) and Good Clinical Practice (GCP) guidelines and with the applicable local regulatory requirements. Moreover, the site will keep all information obtained from the participation in this study confidential unless otherwise agreed in writing.

| Principal Investigator | | |
|---|---|---|
| Print Name | Signature | Date |
| Associate Clinical Operations Mana<br>Valneva Austria GmbH | ger Signature | Date |
| Clinical Strategy Manager<br>Valneva Austria GmbH | Signature | Date |
| Valneva Austria GmbH | CONFIDENTIAL | page 2 / 90 |

#### 2. STUDY PERSONNEL

# Head Clinical Operations Chikungunya Vaccine Development



## Sponsor's Medical / Safety Officer



## **Study Medical Monitor**



## 2.1 Study Organization

The contact details of the organization/individuals involved in the study (e.g.; investigator(s), Sponsor's representative(s), laboratories, oversight committees [including institutional review boards (IRBs), as applicable] will be maintained by the Sponsor and provided to the Investigator.

IND No: 17854

## 3. SERIOUS ADVERSE EVENT REPORTING

The Investigator will comply with applicable laws/requirements for reporting serious adverse events (SAEs) to the IRB. For information on the definition and assessment of adverse events (AEs), refer to Section 17.1.

All SAEs should be reported on the SAE Report Form to the PRA Safety Desk by fax or email within 24 hours after the Investigator has become aware of the event. Under certain circumstances the initial notification could be done by phone, but nevertheless a written SAE Report Form has to be submitted within 24 hours to:

| PRA Safety Desk |
|-----------------|
| Fax: |
| Email: |
| Safety Hotline: |

#### 4. ADVERSE EVENTS OF SPECIAL INTEREST REPORTING

The Investigator will comply with requirements set forth in this protocol for reporting adverse events of special interest (AESIs). For information on the definition and assessment of adverse events of special interest (AESIs), refer to Section 17.1.3.

All AESIs should be reported on the AESI Report Form to the PRA Safety Desk by fax or email within 48 hours after the Investigator has become aware of the event. Under certain circumstances the initial notification could be done by phone, but nevertheless a written AESI Report Form has to be submitted within 48 hours to:

| PRA Safety Desk |
|-----------------|
| Fax: |
| Email: |
| Safety Hotline: |

#### 5. PREGNANCY REPORTING

The Investigator will comply with applicable laws/requirements for reporting pregnancies to the IRB. For information on the definition and assessment of pregnancies, refer to Section 13.4.

All Pregnancies\* should be reported on the Pregnancy Report Form to the PRA Safety Desk by fax or email <u>within 24 hours</u> after the Investigator has become aware of the event.



\* A pregnancy is not considered an SAE. If a seriousness criterion applies in addition to the pregnancy (e.g. hospitalization, congenital anomaly/birth defect) the pregnancy qualifies as an SAE. In such case a Pregnancy Report Form **and** an SAE Report Form have to be filled out.

## 6. STUDY CHANGES IN RESPONSE TO SARS-COV2 PANDEMIC

The study Sponsor will continuously monitor and evaluate the development of the COVID-19 pandemic in the area of study sites to determine if any measures need to be implemented to mitigate undue risks to the subjects or in response to local governmental recommendations. Such measures may include, temporarily halting further recruitment, switching in-person visits to phone calls, or employing mobile teams to collect serum samples. Any measure would be communicated to the relevant Competent Authority and Institutional Review Board and documented in the CSR. For information on COVID-19 management refer to Section 10.6.

#### 7. CLINICAL STUDY SYNOPSIS

| INVESTIGATIONAL PRODUCT, DOSAGE AND MODE OF ADMINISTRATION | |
|---|---|
| Title | A RANDOMIZED, DOUBLE-BLINDED PHASE 3 STUDY TO DEMONSTRATE LOT-TO-LOT CONSISTENCY OF THREE LOTS OF A LIVE-ATTENUATED CHIKUNGUNYA VIRUS VACCINE CANDIDATE (VLA1553) IN HEALTHY ADULTS AGED 18 TO 45 YEARS |
| Name of Investigational Medicinal Product (IMP) | Live-attenuated Chikungunya (CHIKV) vaccine (VLA1553) |
| Name(s) of Active Ingredient(s) | Live-attenuated CHIKV vaccine strain based on the La Reunion strain (LR-CHIKV clone LR2006-OPY1) of East Central South African (ECSA) genotype (del5nsP3) |

VLA1553 is a live-attenuated chikungunya virus (CHIKV) vaccine candidate designed for active immunization for the prevention of disease caused by CHIKV. The candidate vaccine is intended to prevent CHIKV infections in the general population living in endemic regions, as well as to serve as a prophylactic measure for travelers to epidemic areas or areas at risk for an upcoming outbreak or ongoing endemic transmission. The replicating CHIKV vaccine comprises a large deletion of 60 amino acids in the nsP3 gene (del5nsP3) encoding the non-structural replicase complex protein nsP3, which leads to attenuation of the virus *in vivo*.

In this Phase 3 study, three Lots of VLA1553 (target 1x 10E4 TCID<sub>50</sub> per 0.5 mL dose) will be evaluated for immunogenicity to demonstrate manufacturing consistency, as well as for safety. VLA1553 will be administered intramuscularly (i.m.) into the deltoid muscle as a single-shot immunization on Day 1. Subjects will be followed for safety, immunogenicity and antibody persistence up to 6 months. The vaccine presents in a lyophilized dosage form.

CHIKV is a small spherical RNA virus and a member of the Alphavirus genus in the family *Togaviridae*. The arthropod-borne virus is closely related to other viruses in Africa, South America and Australia that cause similar signs and symptoms such as Ross River virus, Mayaro-virus or o'nyong-nyong-virus. The virus is vectored by the daytime-biting *Aedes aegypti* mosquito, which also transmits yellow fever, Zika and dengue viruses. CHIKV can also be transmitted by *Aedes albopictus* mosquitoes, a more cold-tolerant mosquito that could result in the spread of chikungunya to more temperate areas of the world such as Italy and France.

CHIKV has been reported in over 100 countries with more than 2.2 million suspected cases reported to the Pan American Health Organization (PAHO) in the Americas alone. CHIKV epidemics are explosive and rapidly moving, but not predictable.

An infection with CHIKV results in chronic and incapacitating arthralgia affecting all gender and age groups accompanied by an acute febrile disease with headache, muscle pain, and skin rashes. The severe, often debilitating joint pain in infected patients can persist for years, especially in adults. Individuals who are at higher risk of more serious complications include infants, the elderly and individuals with chronic medical conditions. Currently, neither specific antiviral treatment nor a vaccine is available to prevent CHIKV infection. Prevention against CHIKV infection is therefore limited to non-treatment interventions such as the deployment of insecticides, wearing long sleeves and pants and

| repellants, and other means to restrict exposure to vector mosquitos. | |
|---|---|
| CLINICAL CONDITIO | N(S)/INDICATION(S) |
| Active immunization fo | r the prevention of disease caused by CHIKV |
| STUDY PHASE | STUDY PHASE Phase 3 |
| PLANNED STUDY PE | RIOD |
| Initiation | Q1/2021 |
| Duration | The overall study duration (First Subject In – Last Subject Out) is estimated to be approximately 8 months. |
| | Individual subject participation is approximately 7 months from enrollment to study completion unless prematurely discontinued. |
| Completion | Part A (Visit 3, Day 29): planned Q1 / 2021 |
| | Part B (Visit 5, Month 6): planned Q4 / 2021 |
| | Part A analysis will be performed on Day 29 and will comprise the primary endpoint. Part B final analysis will be performed once the last subject has completed Month 6 (Visit 5). |

## **STUDY OBJECTIVES**

## **Primary Objective**

➤ To demonstrate Lot-to-Lot manufacturing consistency of a live-attenuated CHIKV vaccine candidate (VLA1553) 28 days following vaccination in a healthy population aged 18 to 45 years after a single immunization.

## **Secondary Objective**

> To evaluate immunogenicity and safety of VLA1553 up to 180 days following vaccination in a healthy population aged 18 to 45 years after a single immunization.

| STUDY DESIGN | IGN |
|---|---|
| Investigator and sites | Multicenter study. The study will be conducted at approximately four study sites in the U.S. |
| Study participants | A total of approximately 402 healthy subjects aged 18 to 45 years will be enrolled (i.e. ICF signed) and randomized 1:1:1 to receive one of three lots of VLA1553. |
| Study Type | Immunogenicity and Safety |
| Vaccine Type | Live-attenuated CHIKV in a lyophilized formulation |

| ١ | /aln | eva | Αı | ictria | Gmh | Ή |
|---|------|-----|----|--------|-----|---|

| Control Type | Active Control – Lot-to-Lot consistency Prevention |
|---|---|
| Study Indication Type | |
| Blinding Scheme | Blinded (double-blind, i.e. the subject as well as all study site staff/ Investigator/ Sponsor remain blinded to treatment allocation) |

## Study Design

This is a prospective, randomized, double-blinded, multicenter Phase 3 clinical study investigating three lots of VLA1553 at the final dose (target  $1x\ 10E4\ TCID_{50}$  per  $0.5\ mL$ ). Overall, 402 subjects will be enrolled into the study, 134 subjects per VLA1553 Lot (**Table 1**).

Subjects will be block-randomized in a 1:1:1 ratio into the three study arms to receive either of three Lots of VLA1553 as a single i.m. vaccination on Day 1 (Visit 1).

All subjects will be asked to return to the study site at Day 8 (Visit 2), Day 29 (Visit 3), Day 85 (Visit 4) and Month 6 (Day 180, Visit 5) for immunogenicity sampling. Safety data collection will capture solicited AEs until Day 11 and unsolicited AEs up to Day 180 (Month 6, Visit 5) from all subjects. AESIs will be captured 2 to 21 days post-vaccination. Subjects presenting with acute arthralgia within this time period will be followed-up until resolution and monitored for recurrences until the end of the study. SAEs will also be assessed until the end of the study in all subjects (Month 6, Visit 5).

Table 1 below illustrates the individual subject distribution.

| Table 1. Subject Distribution | | | | | |
|---|---|---|---|---|---|
| Study<br>Arm | Vaccine | Cohort | Number of subjects (n) | Target Dose<br>(TCID <sub>50</sub> /dose) | Injection<br>Volume (mL) |
| 1 | VLA1553 | Lot 1 | 134 | 1x 10E4 TCID <sub>50</sub><br>per 0.5 mL | 0.5 |
| 2 | VLA1553 | Lot 2 | 134 | | 0.5 |
| 3 | VLA1553 | Lot 3 | 134 | | 0.5 |
| | | Total N: | 402 | | |

The clinical study design is displayed in the Figure 1 below.



#### STUDY ENDPOINTS

## **Primary Endpoint**

## Immunogenicity:

Geometric mean titer (GMT) of CHIKV-specific neutralizing antibodies as determined by microneutralization (μPRNT) assay on Day 29 post-vaccination in subjects who tested negative for CHIKV antibodies at baseline.

## **Secondary Endpoints**

## Immunogenicity:

- Immune response as measured by CHIKV-specific neutralizing antibody titers on Day 8, Day 85 and Month 6 post-vaccination as determined by µPRNT assay;
- Proportion of subjects with seroprotective levels defined as for baseline negative subjects at Days 8, 29, 85 and Month 6 post- vaccination by μPRNT assay;
- Proportion of subjects with seroconversion<sup>i</sup> at Day 29, and Month 6 as determined by μPRNT assay;
- Fold increase of CHIKV-specific neutralizing antibody titers determined by μPRNT assay at Days 8, 29, 85 and Month 6 post-vaccination as compared to baseline;
- Proportion of subjects reaching an at least 4-fold, 8-fold, 16-fold or 64-fold increase in CHIKV-specific neutralizing antibody titer compared to baseline as measured by μPRNT assay.

#### Safety:

- Frequency and severity of solicited injection site and systemic reactions within 10 days post-vaccination;
- Frequency and severity of unsolicited adverse events (AEs) within 28 days post-vaccination;
- Frequency and severity of any adverse event (AE) during the entire study period;

i Seroconversion defined as CHIKV-specific neutralizing antibody titer of for baseline negative subjects and for baseline positive subjects.

- Frequency and severity of any serious adverse event (SAE) during the entire study period;
- Frequency and severity of any adverse event of special interest (AESI) within 2 to 21 days post-vaccination.

#### **CRITERIA FOR INCLUSION / EXCLUSION**

Approximately 402 adults of either gender, who satisfy the inclusion and exclusion criteria listed below will be invited to participate in the study.

#### **Inclusion Criteria**

Subjects who meet ALL of the following criteria are eligible for this study:

- 1. Subject is 18 to 45<sup>ii</sup> years of age on the Day of screening (Visit 0);
- 2. Subject has an understanding of the study and its procedures, agrees to its provisions, and voluntarily gives written informed consent prior to any study-related procedures;
- 3. Subject is generally healthy<sup>iii</sup> as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests;
- 4. If subject is of childbearing potential:
  - a) Subject has practiced an adequate method of contraception (see below) during the 30 days before screening (Visit 0);
  - b) Subject has a negative serum or urine pregnancy test at screening (Visit 0) or Visit 1, respectively;
  - c) Subject agrees to employ adequate birth control measures for the first three months post-vaccination (i.e. until Day 85, Visit 4). This includes one of the following measures:
    - Hormonal contraceptives (e.g. implants, birth control pills, patches);
    - Intrauterine hormone-release systems and intrauterine device;
    - Barrier type of birth control measure (e.g. diaphragms, cervical caps);
    - Vasectomy in the male sex partner ≥ 3 months prior to first vaccination:
    - Sexual abstinence:
    - Same sex relationships;
    - Condoms when used in combination with any of the female contraceptive measures outlined above<sup>iv</sup>.

#### **Exclusion Criteria**

Subjects who meet ANY of the following criteria are NOT eligible for this study:

Subject has had a CHIKV infection in the past (self-reported), including suspected CHIKV infection; is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical study involving an investigational

From the 18th birthday until the last day before the 46th birthday.

Subjects are considered **generally healthy** if (1) any chronic illness/condition, e.g. hypertension, type 2 diabetes mellitus, or hyperlipidemia is stable and well-controlled on therapy for the past 6 months, and (2) they do not have a disease that is identified as an exclusion criterion.

iv Condoms are not to be used as a sole means of contraception.

#### CHIKV vaccine;

- 2. Subject has an acute or recent infection (and who is not symptom-free in the week prior to the Screening Visit (Visit 0);
- 3. Subject tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
- 4. Subject has received another live virus vaccine within 28 days or inactivated vaccine within 14 days prior to vaccination in this study or plans to receive a vaccine within 28 days or 14 days after vaccination, respectively;
- 5. Subject has abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the study based on his/her judgement;
- 6. Subject has a medical history of or currently has acute or progressive, unstable or uncontrolled clinical conditions (e.g. cardiovascular, respiratory, neurologic, psychiatric, or rheumatologic conditions) that poses a risk for participation in the study, based on Investigators clinical judgement. Examples include individuals with poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment, or presence of high-risk comorbidities (e.g. significant cardiopulmonary disease);
- 7. Subject has a history of immune-mediated or clinically relevant arthritis/arthralgia;
- 8. Subject has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the subject may be enrolled. A history of hematologic malignancy is a permanent exclusion. Subjects with a history of skin cancer must not be vaccinated at the previous tumor site;
- 9. Subject has a known or suspected defect of the immune system, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day within 4 weeks prior to study entry, radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous 3 years; topical and inhaled steroids are allowed.
- 10. Subject has a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications):
- 11. Subject presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws;
- 12. Subject is pregnant (positive serum or urine pregnancy test at screening or Visit 1, respectively), has plans to become pregnant during the first three months post-vaccination or lactating at the time of enrollment;
- 13. Subject has donated blood, blood fractions or plasma within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or plans to donate blood or use blood products until Day 180 of the study;
- 14. Subject has a rash, dermatological condition or tattoos that would, in the opinion of the

Investigator, interfere with injection site reaction rating;

- 15. Subject has a known or suspected problem with alcohol or drug abuse as determined by the Investigator;
- 16. Subject has any condition that, in the opinion of the Investigator, may compromise the subjects well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
- 17. Subject is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
- 18. Subject has participated in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study;
- 19. Subject is a member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

## **Delay Criteria**

Vaccination will be delayed if:

- 1. Subject has an acute febrile infection within 72 hours prior to vaccination or oral temperature greater than or equal 38.0 °C/ 100.4 °F on the day of vaccination (subject may be rescheduled within the screening visit window until subject has completed 72 hours of no fever);
- 2. Subject has received antipyretics within 4 hours prior to the scheduled time of vaccination (subject may be rescheduled within the screening visit window).
- 3. Subject has received any live or inactivated vaccine within 28 days or 14 days prior to vaccination, respectively.

In addition, for a rescheduled vaccination all inclusion and none of the exclusion criteria must be met; in case not all of these criteria are met, the subject will be excluded from the study.

The rescheduled visit should be within the specified time window for the vaccination visit. In case the time window for the rescheduled visit cannot be met, the subject might be invited for a re-screening.

Subjects who have been screen failed under protocol version 2.0 due to the site not receiving the subjects CHIKV-serostatus from the testing laboratory within the 28 day screening window can be asked back for re-screening. All eligibility tests will again be performed with the exception of the CHIKV-serostatus test<sup>v</sup>.

Moreover, re-screening will not be allowed for subjects who screen fail to other reasons, such as

Valneva Austria GmbH

CONFIDENTIAL

<sup>&</sup>lt;sup>v</sup> The original CHIKV result from the sample taken at the initial screening visit will be valid for up to 60 days from sample collection.

inclusion/exclusion criteria.

#### STATISTICAL ANALYSIS

### **Sample Size Justification**

The sample size is selected to allow for a demonstration of Lot-to-Lot consistency based on the primary endpoint, CHIKV-specific neutralizing antibody titers as determined by microneutralization ( $\mu$ PRNT) assay on Day 29 post-vaccination. The primary analysis will demonstrate equivalence between the three treatment groups based on a comparison of GMTs.

402 randomized subjects (i.e. 134 per batch) will ensure that the three pair-wise comparisons have an overall power of approximately 90% based on a two-sided significance level of 5%, an assumed SD of 0.32 (on a log10 scale), and acceptance margins of for the GMT ratios, while correcting for an assumed drop-out rate of 10%, 5% of subjects with major protocol deviations and 2% of subjects expected to be baseline positive for CHIKV.

#### **Statistical Methods**

The primary immunogenicity analysis will be a comparison of the GMTs in the per-protocol population (PP) who tested negative for CHIKV antibodies at baseline, analysis set between the VLA1553 Lots 1, 2 and 3 at Day 29 (i.e. 28 days post-vaccination) by ANOVA (factor Lot, covariate study site). GMTs and GMT ratios will be estimated taking the anti-log of the resulting point estimates for the least squares means, least squares means differences and the corresponding 2-sided 95% CIs. If the three resulting confidence intervals obtained from the pair-wise comparisons lie within the interval equivalence of the three lots will be postulated. A statistical analysis plan will be prepared which will detail which immunogenicity analyses will be repeated on the full analysis set.

Secondary immunogenicity analysis will include the comparison of the GMTs between the three Lots at Day 8, Day 85 and Month 6 post-vaccination by ANOVA (factor Lot and covariate study site), two-sided 95% confidence intervals will be calculated for the GMT; GMFls will be analyzed as outlined for GMTs. In addition, the seroprotection and seroconversion rates for various study days, and when applying other threshold titers for defining seroconversion or seroprotection thresholds will be compared between the treatment groups by Fisher's exact test and 95% confidence intervals will be calculated.

All subjects entered into the study, who receive the single vaccination, will be included in the safety analysis.

Safety tabulations will generally be provided separately for solicited AEs and unsolicited AEs, and for both types of AEs combined. 95% confidence intervals according to Altman will generally be provided for all AE rates and differences between the three Lots will be assessed for significance using Fisher's exact test.

The number and percentage of subjects with any AE, any solicited AE, unsolicited AE, any related

unsolicited AE, any related severe AE, any SAEs, any related SAEs, any AESI, any related AESI, any medically attended AE, any AE leading to withdrawal from study, and any AE occurring at a frequency of at least 10% and at least 1% in at least one study arm, up to Day 29, and up to Month 6, will be presented for each Lot overall and by system organ class/ preferred term.

## **Data Analysis**

The following data analyses will be performed:

- Part A includes immunogenicity and safety data after all subjects have completed Visit 3 (Day 29);
- Part B includes immunogenicity and safety data after all subjects have completed Visit 5 (Month 6).

Individual study parts will be analyzed sequentially.

## **Final Report**

The Part A analysis will be performed once the last subject has completed the study Visit 3 (Day 29). Part B analysis will be performed once the last subject has completed the study Visit 5, i.e. (Month 6), respectively. Part A will be unblinded but the blind will be maintained for study sites.

# **8. TABLE OF CONTENTS**

| | PROTOCOL SIGNATURE PAGE | |
|---|---|---|
| 2. | STUDY PERSONNEL | _ |
| ^ | 2.1 Study Organization | |
| ა.<br>⊿ | SERIOUS ADVERSE EVENT REPORTINGADVERSE EVENTS OF SPECIAL INTEREST REPORTING | 4 |
| 5. | PREGNANCY REPORTING | 6 |
| 6. | STUDY CHANGES IN RESPONSE TO SARS-COV2 PANDEMIC | 7 |
| | TABLE OF CONTENTS | |
| | LIST OF ABBREVIATIONS | |
| | ). INTRODUCTION | |
| | 10.1 Valneva's Candidate Vaccine | .24 |
| | 10.2 Clinical Condition/Indication | .24 |
| | 10.2.1 Transmission, Disease and Diagnosis | .24 |
| | 10.2.2 Prospects for Vaccine Development | .25 |
| | 10.3 Findings from Non-clinical and Clinical Studies | .26 |
| | 10.3.1 Non-clinical Summary | .26 |
| | 10.3.2 Clinical Summary | .28 |
| | 10.4 Study Rationale and Justification for Dosage and Study Design | .30 |
| | 10.4.1 Selection of Study Population | .30 |
| | 10.4.2 Selection of Seroprotective Threshold | .30 |
| | 10.5 Evaluation of Anticipated Risks and Benefits of the Investigational Product(s) to Humar Subjects | |
| | 10.5.1 Possible Benefits for Subject | |
| | 10.5.2 Possible Benefits for Society | .31 |
| | 10.5.3 Possible Risks / Inconveniences for the Subject | .32 |
| | 10.6 COVID-19 Management | .33 |
| 11 | . STUDY PURPOSE AND OBJECTIVES | 34 |
| | 11.1 Study Purpose | .34 |
| | 11.2 Primary Objective | .34 |
| | 11.3 Secondary Objective | .34 |
| 12 | 2. STUDY DESIGN | 35 |
| | 12.1 Overall Study Design | .35 |
| | 12.2 Study Duration | .36 |
| | 12.3 Study Endpoints | .36 |
| | 12.3.1 Primary Endpoint | .36 |
| | 12.3.2 Secondary Endpoints | .36 |
| | 12.4 Randomization and Blinding | .37 |

| 12.4.1 Blinding Process | 38 |
|----------------------------------------------------------------------|----|
| 12.4.2 Unblinding | 38 |
| 12.5 Study Termination - Study Stopping Rules | 38 |
| 13. SUBJECT SELECTION, WITHDRAWAL AND DISCONTINUATION | |
| 13.1 Inclusion Criteria | 39 |
| 13.2 Exclusion Criteria | 39 |
| 13.3 Delay Criteria for Vaccination | 41 |
| 13.4 Pregnancy Testing and Birth Control | 42 |
| 13.5 Subject Withdrawal or Discontinuation | 43 |
| 14. INVESTIGATIONAL MEDICINAL PRODUCT | 45 |
| 14.1 Description of VLA1553 | 45 |
| 14.2 IMP Packaging, Labeling, and Storage | |
| 14.2.1 VLA1553 Packaging | 45 |
| 14.2.2 IMP Labeling | 46 |
| 14.2.3 IMP Storage | 46 |
| 14.2.4 Dispensing and Accountability of IMP | |
| 15. STUDY PROCEDURES | |
| 15.1 Informed Consent and Enrollment | |
| 15.2 Subject Identification Code | |
| 15.3 Investigational Treatment | |
| 15.3.1 Description of Treatment | |
| 15.3.2 Vaccine Preparation and Administration | |
| 15.3.3 Post- Vaccination Observation | |
| 15.4 Screening and Study Visits | |
| 15.4.1 Part A | |
| 15.4.2 Part B | |
| 15.4.3 Unscheduled Visit | |
| 15.4.4 Early Termination Visit | |
| 15.5 Procedures for Monitoring Subject Compliance | |
| 16. ASSESSMENT OF IMMUNOGENICITY | |
| 16.1 Determination of vaccine-induced neutralizing antibody response | |
| 16.2 Additional Testing Procedures | |
| 17. ASSESSMENT OF SAFETY | |
| 17.1 Adverse Events | |
| 17.1.1 Adverse Events | |
| 17.1.3 Adverse Events of Special Interest | |
| 11.1.0 / NOVOIDO EVOIRO OF OPONOR INTEREST | |

| 17.1.4 Medically-Attended Adverse Event | 56 |
|-------------------------------------------------------------------|----|
| 17.1.5 Preexisting Diseases | 56 |
| 17.1.6 Untoward Medical Occurrences Not Considered Adverse Events | 56 |
| 17.2 Collection, Documentation and Assessment of Adverse Events | 56 |
| 17.2.1 Unsolicited Adverse Events | 56 |
| 17.2.1.1 Severity | 57 |
| 17.2.1.2 Causality | 57 |
| 17.2.1.3 Assessment and Outcome of Adverse Events | 58 |
| 17.2.2 Solicited Adverse Events | 59 |
| 17.2.2.1 Injection Site Reaction – Measurement and Evaluation | 59 |
| 17.2.2.2 Systemic Reactions – Measurement and Evaluation | 60 |
| 17.2.2.3 Body Temperature Measurement | 61 |
| 17.3 Study eQuestionnaires | 62 |
| 17.4 Medical, Medication, and Non-Drug Therapy History | 63 |
| 17.4.1 Medical history | 63 |
| 17.4.2 Concomitant Medications and Non-Drug Therapies | 64 |
| 17.5 Vital Signs | 65 |
| 17.6 Physical Examinations | 65 |
| 17.7 Clinical Laboratory Parameters | 66 |
| 17.7.1 Safety Sample | |
| 17.7.2 CHIKV Screening | |
| 17.7.3 COVID-19 Sample | 67 |
| 17.7.4 Baseline Sample | 67 |
| 17.7.5 Assessment of Laboratory Values | 67 |
| 17.8 Viremia | 68 |
| 17.9 Adverse Events of Special Interest (AESI) | 68 |
| 17.10 Adverse Event Reporting Procedures | 69 |
| 17.10.1 Serious Adverse Event | 69 |
| 17.10.2 Adverse Events of Special Interest (AESI) | 70 |
| 17.10.3 Pregnancy | 70 |
| 17.11 Safety Monitoring | 71 |
| 17.11.1 Data Safety Monitoring Board | 71 |
| 17.11.2 Sponsor | 72 |
| 17.11.3 Investigator | 72 |
| 18. STATISTICS | 73 |
| 18.1 Sample Size Justification | 73 |
| 18.2 Datasets and Analysis Cohorts | 73 |

| 18.3 Handling of Missing, Unused, and Spurious Data | 74 |
|---|---|
| 18.4 Methods of Analysis | 74 |
| 18.4.1 Primary Endpoint | 74 |
| 18.4.2 Secondary Endpoints | 74 |
| 18.4.2.1 Secondary Safety Endpoints | 74 |
| 18.4.2.2 Secondary Immunogenicity Endpoints | 75 |
| 18.5 Planned Data Analysis of the Study | 75 |
| 19. ETHICS AND REGULATORY ASPECTS | 76 |
| 19.1 Compliance Statement | 76 |
| 19.2 Institutional Review Board (IRB) and Regulatory Authorities | 76 |
| 19.3 Subject Information and Informed Consent | 76 |
| 20. QUALITY CONTROL AND QUALITY ASSURANCE | |
| 20.1 Source Data and Records | |
| 20.2 Investigator's Responsibility | 77 |
| 20.3 Training | <b>7</b> 7 |
| 20.4 Monitoring | 78 |
| 20.5 Audit and Inspection | 78 |
| 20.6 Non-compliance with the Protocol / Protocol Deviations from the Protocol | 78 |
| 20.7 Confidentiality of Subject's Data | 78 |
| 21. DATA HANDLING AND RECORD KEEPING | |
| 21.1 Information of Investigators | 78 |
| 21.2 Electronic Case Report Forms (eCRFs) | 79 |
| 21.2.1 Data Recorded Directly on Case Report Forms | |
| 21.2.2 eCRF entries | 79 |
| 21.2.3 Changes to eCRF data | 79 |
| 21.2.4 eCRF Entry Validation | |
| 21.2.5 Data collection | 80 |
| 21.3 Coding of Adverse Events, Drugs and Diseases | 80 |
| 21.4 Investigator File | 80 |
| 21.4.1 Maintenance | |
| 21.4.2 Archiving and Destruction | 80 |
| 21.4.3 Provision of Additional Information | |
| 22. PUBLICATION POLICY | |
| 23. LIABILITIES AND INSURANCE24. SUPPLEMENTS | |
| 24.1 Study Flow Chart | |
| 24.2 Schedule of Study Procedures and Assessments | |

| VLA1553 | Clinical Study Protocol VLA1553-302 Final 3.0<br>IND No: 17854 | 07-Apr-2021 |
|---|---|---|
| 24.3 Toxicity Grading | Scale for Abnormal Laboratory Assessments | 85 |
| 24.4 Guidance on Hai | 87 | |
| 25 REFERENCES | | 80 |

# 9. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|-------------------------------------------|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ANOVA | Analysis of variance |
| ALT | Alanine aminotransferase |
| aPTT | Activated Partial Thromboplastin Time |
| AST | Aspartate aminotransferase |
| BMI | Body Mass Index |
| CDC | Centers of Disease Control and Prevention |
| CHIKV | chikungunya virus |
| CI | Confidence interval |
| CRA | Clinical research associate |
| CRO | Contract Research Organization |
| CRP | C-reactive protein |
| CSR | Clinical Study Report |
| DSMB | Data and Safety Monitoring Board |
| eCRF | electronic Case Report Form |
| e.g. | for example |
| ESR | Erythrocyte sedimentation rate |
| FDA | Food and Drug Administration |
| GMFI | Geometric mean fold increase |
| GMT | Geometric mean titer |
| Hb | Hemoglobin |
| HBsAg | Hepatitis B surface antigen |
| HCV | Hepatitis C virus |
| Hct | Hematocrit |
| HIV | Human immunodeficiency virus |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| i.e. | that is |
| i.m. | Intra - muscular |
| IMP | Investigational medicinal product |

# Clinical Study Protocol VLA1553-302 Final 3.0 IND No: 17854

07-Apr-2021

| Abbreviation | Definition |
|---|---|
| IRB | Intitutional Review Board |
| IXRS | Interactive Voice/Web Response System |
| kDa | kilo Dalton |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mL | Milliliter(s) |
| n.a. | not applicable |
| NT | Neutralization Test |
| NT <sub>50</sub> | Antibody titer at 50% virus neutralization (as determined in Phase 1 microneutralization assay) |
| PCR | Polymerase chain reaction |
| рН | Potential of hydrogen |
| PP | Per-protocol |
| μPRNT | Micro Plaque Reduction Neutralization Test |
| μPRNT <sub>50</sub> | PRNT titer based on a 50% reduction in plaque count |
| RBC | Red blood cells |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| S.C. | subcutaneous |
| SPR | Seroprotection Rate |
| WBC | White blood cell |

#### 10. INTRODUCTION

#### 10.1 Valneva's Candidate Vaccine

Valneva has developed a live-attenuated chikungunya virus (CHIKV) vaccine candidate VLA1553 for the active prevention of chikungunya infection for use in endemic regions and for travelers to epidemic areas or high risk areas. VLA1553 is based on the chikungunya La Reunion strain (LR-CHIKV clone LR2006-OPY1) of East Central South African (ECSA) genotype and is characterized by a genetically-engineered 60 amino acid deletion in its nsP3 viral replicase complex gene which leads to an attenuation of the virus *in vivo*. VLA1553 is genetically stable and passaged three times on African green monkey kidney (VERO) cells and contains no adjuvant. VLA1553 is intended to facilitate a rapid development of a protective antibody titer.

VLA1553 investigation was designated as a fast track development program by the United States (US) Food and Drug Administration (FDA) in 2019.

For further details please refer to the Investigator's Brochure.

#### 10.2 Clinical Condition/Indication

#### 10.2.1 Transmission, Disease and Diagnosis

CHIKV is a mosquito-borne virus which was first isolated in 1953, during an epidemic of polyarthralgia in Tanzania (Robinson 1955). The word 'chikungunya' means 'that which bends up' in Swahili, in reference to the stooped posture of patients afflicted with the severe joint pain associated with this disease. Since its first isolation CHIKV was found to occasionally cause smaller outbreaks during the following decades in Africa, India, the Indian Ocean Islands, and Southeast Asia (Suhrbier, Jaffar-Bandjee et al. 2012; Simon, Javelle et al. 2015).

Within the human population, CHIKV is maintained by a human-mosquito-human transmission probably following a dengue-like model characterized by the absence of an animal reservoir and the ability to spread rapidly among human beings via domestic and peridomestic mosquitoes (Pialoux, Gauzere et al. 2007; Her, Kam et al. 2009). CHIKV was typically transmitted only by *Aedes aegypti* mosquitos, however coinciding with an adaptation enabling unusually efficient transmission by *Aedes albopictus* mosquitos, the virus re-merged in 2004 and rapidly spread over Africa, Asia and locally also in Europe (Delisle, Rousseau et al. 2015). More recently CHIKV also has spread across the Americas with millions of people becoming infected (Rezza, Weaver et al. 2019).

CHIKV is an enveloped alphavirus of the family *Togaviridae*. It carries a single-stranded positive sense genomic RNA of around 12 kb containing two open reading frames that

encode four nonstructural replicase proteins (nsP1-4) and a structural polyprotein consisting of the capsid protein (C) and the envelope proteins (E3-E2-6K-E1), respectively. The replicase complex serves two functions: it replicates the genomic RNA for incorporation into new virus particles and it also has transcriptase activity to produce a mRNA from a subgenomic promoter that encodes the structural proteins (Simizu, Yamamoto et al. 1984). Mature virions that bud from the plasma membrane of infected cells carry 240 copies of E2-E1 glycoproteins arranged into 80 heterotrimeric spike complexes. The E2 protein is the receptor-binding moiety, whereas the E1 protein is involved in fusion of the virion envelope with the target cell endosomal membrane (Voss, Vaney et al. 2010). Accordingly, it is the spike complex and in particular the E2 envelope protein that is the target for neutralizing antibodies.

An infection with CHIKV results in chronic and incapacitating arthralgia affecting all gender and age groups (Couderc, Khandoudi et al. 2009; Suhrbier, Jaffar-Bandjee et al. 2012; Simon, Javelle et al. 2015). CHIKV clinical symptoms are presented in three stages that differ in clinical features and treatment. During the acute stage, clinical symptoms manifest with common features such as fever, transient rash and multiple arthralgia/arthritis episodes. This is followed by a multi-morbid post-acute and chronic stage characterized by persisting rheumatic symptoms up to months and years after infection and impaired quality-of-life (Marimoutou, Ferraro et al. 2015; Simon, Javelle et al. 2015). Symptoms of CHIKV disease usually appear 4–7 days post-infection and include rapid onset of fever, viremia, severe joint pain, recurring mild joint pain, maculopapular rash, and may lead to death (Simon, Javelle et al. 2015).

Currently, neither specific antiviral treatment nor a vaccine is available to prevent CHIKV infection. Prevention against CHIKV infection is therefore limited to non-treatment interventions such as the employment of insecticides, wearing long sleeves and pants and repellents, and other means to restrict exposure to vector mosquitos. The treatment of CHIKV disease is mainly supportive such as bed rest, adequate fluids, and symptomatic relief by using analgesics, antipyretics like paracetamol, or anti-inflammatory drugs like ibuprofen and naproxen for the control of fever and joint pain. Persons who have persistent joint pain may require analgesic or long-term anti-inflammatory therapy (Simon, Javelle et al. 2015).

For detailed information on the disease and epidemiology please refer to the Investigator's Brochure.

#### 10.2.2 Prospects for Vaccine Development

A number of CHIKV vaccine candidates is currently under pre-clinical and clinical development, ranging from inactivated whole virus vaccine compositions, over virus-like-particle approaches to RNA and DNA vaccine candidates (Schrauf et al. 2020).

A former CHIKV vaccine candidate was a serially passaged, live-attenuated CHIKV vaccine (TSI-GSD-218 or 181/clone 25) developed by the Walter Reed Army Institute of Research (WRAIR, US). The TSI-GSD-218 CHIKV isolate was derived from a patient during the Thailand outbreak in 1962 and was subsequently serially passaged on human lung cell cultures. The live-attenuated vaccine candidate was investigated in numerous Phase 1 and Phase 2 trials with a dose of 3x10<sup>4</sup> PFUs/mL. The WRAIR vaccine was administered i.m. as well as subcutaneous (s.c.) as a single vaccination offering long-term protection (McClain, Pittman et al. 1998 and Edelman, Tacket et al. 2000). However, clinical development efforts were terminated in 1998 (Hoke, Pace-Templeton et al. 2012).

In addition, a measles-virus-based CHIKV vaccine developed by Themis, AT, has completed Phase 1 and 2 studies. Published results of a Phase 2 clinical trial investigating two immunizations of escalating dose levels at four sites in Austria and Germany showed that the vaccine was found to be safe and well-tolerated with a good immunogenicity profile (Ramsauer, Schwameis et al. 2015, Reisinger et al. 2018).

Furthermore, the National Institutes of Allergy and Infectious Disease (NIAID), later acquired by PaxVax, now Emergent BioSolutions, developed a Virus-like particle (VLP) vaccine for prophylaxis of CHIKV. Fist-in-human and Phase 2 studies demonstrated in non-endemic and endemic regions of the Caribbean that the VLP vaccine candidate is safe, well-tolerated and immunogenic after two vaccinations supporting Phase 3 entry (Chen et al. 2020; Chang et al. 2014).

With the increase of international travel in the past years and the spread of potential vectors, infections caused by CHIKV are likely to expand on a global scale and may result in overlapping regions of endemicity (Hochedez, Jaureguiberry et al. 2006). Consequently, morbidity due to this virus is a serious threat to global health, and CHIKV has been listed as a priority pathogen by the National Institutes of Allergy and Infectious Disease (NIAID) in the United States (Suhrbier, Jaffar-Bandjee et al. 2012; Simon, Javelle et al. 2015; NIAID October 26, 2016) and raises an urgent demand for efficient prophylaxis, providing a strong justification for the development of a vaccine.

#### 10.3 Findings from Non-clinical and Clinical Studies

#### 10.3.1 Non-clinical Summary

The safety, immunogenicity and protective potency of the CHIKV vaccine candidate VLA1553 have been assessed in numerous non-clinical studies.

The non-clinical development program has focused on the establishment of a small animal as well as non-human primate (NHP) model allowing for the evaluation of the CHIKV candidate vaccine with respect to safety and efficacy, i.e. immunogenicity and protection (Hallengärd et al. 2014). To this end, mouse models have been investigated and were shown to be permissive for infection with a wild-type (wt) CHIKV isolate, LR2006 OPY-1.

Thus, infection of mice with wt CHIKV was shown to cause significant viremia, a major sign also in humans (Couderc and Lecuit 2009). In addition, NHPs serve as excellent animal models for understanding CHIKV pathogenesis as they are a natural amplification host for CHIKV and share significant genetic and physiological homology with humans. CHIKV infection in NHPs results in acute fever, rash, viremia and the production of CHIKV-specific neutralizing antibodies, type I interferon and pro-inflammatory cytokines. CHIKV establishes a persistent infection in NHPs, particularly in cynomolgus macaques (Broeckel, Haese et al. 2015).

Valneva's pre-clinical data package generated with the CHIKV vaccine candidate demonstrates that a single shot of the CHIKV del5nsP3 vaccine/VLA1553:

- ➤ is highly immunogenic and induces a strong and long lasting neutralizing antibody response in a mouse and NHP model;
- protects NHPs from a high-dose wt CHIKV challenge;
- > causes no clinical manifestations typically associated with wt CHIKV infections in the NHP model;
- shows a delayed and strongly reduced viremia as compared to wt CHIKV infection in a mouse and NHP model;
- > shows strongly reduced cytokine production compared to wt CHIKV infection;
- > shows a more sporadic, transient and lower dissemination in tissues of VLA1553;
- immunized NHPs compared to wt CHIKV infected NHPs;
- > confirms the stability of the virus del5nsP3 attenuation in humans post-vaccination;
- ➤ is able to protect NHPs from CHIKV infection based on passive transfer of human immune sera to NHPs followed by wt CHIKV challenge and
- > shows a negligible risk of VLA1553 virus transmission from vaccinated to non-vaccinated humans by mosquitoes.

An overview of further non-clinical studies can be found in **Table 2** below.

Table 2. Non-clinical Studies with VLA1553

| Study | Species | Summary |
|---|---|---|
| Repeat-Dose Toxicity | Rabbits<br>(New Zealand<br>Whites) | Upon two high dose vaccinations at a two week interval, all findings were transient and resolved within the 30 days recovery period; No adverse findings. |
| Persistence of infection and biodistribution | NHPs<br>(Cynomolgus<br>macaques) | <ul> <li>VLA1553 replication in blood was 3 logs lower than replication of wt CHIKV;</li> <li>shedding of VLA1553 in saliva and vaginal fluids was much lower than wt CHIKV;</li> <li>in cerebrospinal fluid, synovial fluid and urine, no shedding of VLA1553 nor wt CHIKV was detected;</li> <li>VLA1553 dissemination in tissues, when detected, was more sporadic, transient and lower than observed for wild-type CHIKV;</li> <li>VLA1553 was not detected in joints and muscles.</li> </ul> |
| Mosquito Transmission Study | Mosquitos<br>(Aedes albopictus) | Probability of mosquitoes transmitting VLA1553 virus from a human vaccinated with the vaccine appears to be minisculy low (threshold titer of |
| Passive transfer in NHPs using human serum from VLA1553-101 | NHPs<br>(Cynomolgus<br>macaques) | After vaccination with VLA1553 is proposed as a titer reasonably likely to predict protection. |

For further details please refer to the Investigator's Brochure.

## 10.3.2 Clinical Summary

The first clinical study with Valneva's live-attenuated vaccine candidate was initiated with first-subject-in on 05 March 2018 in the U.S. and was designed as randomized, observerblinded, multicenter Phase 1 dose-escalation study (VLA1553-101) assessing both safety and immunogenicity. The study has been conducted in healthy male and female (of nonchildbearing potential) volunteers aged 18 to 45 years, who are unlikely to have had a natural infection with CHIKV (naïve population). Three escalating dose levels of VLA1553 of 3.2x10<sup>3</sup>, 3.2x10<sup>4</sup> or 3.2x10<sup>5</sup> TCID<sub>50</sub>/dose in a liquid formulation (30 subjects in the low and medium and 60 subjects in the high dose group) were investigated after a single immunization in a total of 120 subjects. Dosing was adjusted by injection volume. All subjects returned to the study site at Day 28 and Day 84, Month 6 and at Month 12 for safety and immunogenicity evaluations. Subjects in dose groups L and M were revaccinated ("intrinsic human virus challenge") with the highest dose at Month 12 and followed up for safety and immunogenicity until 28 days after re-vaccination, i.e. until Month 13. Subjects in dose group H were re-randomized 1:1 at Month 6 to receive either a revaccination with the highest dose at this Visit 4 or at Month 12. Subjects were followed up for safety and immunogenicity until 28 days after their respective re-vaccination, i.e. until Month 7 and further continued until Month 12 or Month 13, respectively. Additionally, throughout the study, subjects returned to the study site for safety, including the assessment of viremia, shedding and CHIKV-associated events, as well as immunogenicity evaluations on Days 3, 7 and 14 post-vaccinations. Should a subject present with a positive viremia or shedding sample on Day 14 after vaccination, weekly tests are performed until viremia/shedding were resolved.

Taken together, VLA1553 was well-tolerated in the low and medium dose groups and generally safe in all dose groups after a single vaccination. The low and medium doses of VLA1553 have a superior safety profile (including viremia) compared to the high dose group. No AESIs and no SAEs related to vaccination were reported up to Month 12. The local tolerability profile at all dose levels was considered excellent. Notable systemic AEs included short-term fever, headache and muscle pain. Adverse event rates were significantly lower in the low and medium dose groups compared to the high dose group. Following a re-vaccination ("intrinsic human virus challenge") with the highest dose at Month 6 (Group H2) or Month 12 (Group L, M and H1) vaccines were protected from vaccine induced viremia as indicated by the absence of positive viremia results in plasma, urinary shedding as well as associated adverse events. On Day 14, the GMTs in the Low, Medium and High dose groups were and respectively; with statistically significant differences between the Low and Medium and Low and High dose groups.

VLA1553 showed an excellent immunogenicity profile in all dose groups after a single vaccination. 100% Seroconversion rates (conservatively defined as the proportion of subjects achieving a CHIKV-specific neutralizing antibody titer of were already achieved at Day 14 after the single vaccination in all dose groups and was sustained at 100% until Month 12. 96.3% or more subjects in all dose groups achieved at least a 16-fold increase in antibody titers at Day 28. Mean peak antibody titers at Day 28 ranged from GMT from groups L to H, respectively, with maximum titers at Day 28 reaching Neutralizing antibodies persisted up to a year (GMTs ranging from in Group H2 to in Group M). The absence of an anamnestic response following any re-vaccination demonstrates that a single vaccination of VLA1553 is sufficient to induce sustaining high titer neutralizing antibodies at all dose levels one year after priming characterized by the development of sterilizing immunity ( increase in 94.4 to 100.0% of subjects) in neutralizing antibody titers as compared to titers prior revaccination.

For further information on Study VLA1553-101, please refer to the Investigator's Brochure.

In summary, the medium dose was considered equally safe as the low dose but presented with an improved immunogenicity profile in terms of neutralizing antibody kinetics. Based on these results Valneva selected the medium dose of VLA1553 for further clinical development of the vaccine. Based on this solid and comprehensive clinical data package involving data on approximately 120 subjects, wherein 30 have received the final product as a single vaccination, the inclusion of an "intrinsic human virus challenge" with the potential to generate early data on efficacy and the evidence for a single-dose vaccination

schedule supports the advancement of this chikungunya virus vaccine candidate (VLA1553) to this Phase 3 study responding to the urgent medical need for a prophylactic CHIKV vaccine.

### 10.4 Study Rationale and Justification for Dosage and Study Design

Building on the initial data from the Phase 1 study (study VLA1553-101), this Lot-to-Lot Phase 3 study is designed to demonstrate manufacturing consistency of three manufacturing Lots. Additionally, this Lot-to-Lot study as well as the pivotal Phase 3 study (VLA1553-301) are designed to expand the safety and immunogenicity database of the final dose of VLA1553 administered as a single vaccination. The acceptance margins of were chosen for the calculation of study sample size.

## 10.4.1 Selection of Study Population

A total of approximately 402 healthy subjects of either gender, 18 to 45 years of age, who meet all inclusion criteria and none of the exclusion criteria and provide a written informed consent, will be invited to participate in the study. Subjects who have a history of CHIKV infection, including a suspected CHIKV infection or subjects who are taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection will be excluded. Subjects will be screened for their CHIKV sero-status at study entry, subjects tested positive for CHIK will be excluded from the primary endpoint analysis.

## 10.4.2 Selection of Seroprotective Threshold

| Human immune sera derived from individuals of the Phase 1 clinical study (VLA1553-101) with different titers were passively transferred to NHPs to assess protection from vira replication after challenge with a high dose of wt CHIKV LR2006- OPY1. The challenge dose used for this study PFU) corresponds to a dose that is higher than the dose people may encounter when bitten by a mosquito (Dubrulle et al., 2009). |
|---|
| The study revealed, that the animals were fully protected against viremia by using the highest dose of human immune sera (Day 28, |
| Most importantly, the NHP passive transfer study showed that all human VLA1553-101 serum treated animals with µPRNT <sub>50</sub> titers between prior to challenge were fully protected against CHIKV infection-associated fever or modification of blood parameters. The threshold for protection (lowest observed Day 0 titer at which at least 90% of animals are protected from viremia) was |

When comparing the protection against CHIKV infection provided by the human sera of Day 180 post-immunization with the data of the Day 28 (or Day 14 and 84) sera, our analysis showed there is no significant difference in terms of viremia or protection at the same level of  $\mu PRNT_{50}$  titer prior to challenge.

Based on a FDA request to include a conservative safety margin, a neutralizing antibody titer of termined by µPRNT50 is proposed as a titer reasonably likely to predict protection in humans and is therefore an agreed surrogate endpoint to support accelerated approval.

# 10.5 Evaluation of Anticipated Risks and Benefits of the Investigational Product(s) to Human Subjects

## 10.5.1 Possible Benefits for Subject

The benefit of participation for the subjects in this study is the possible formation of antibodies against CHIKV after vaccination with the VLA1553 candidate vaccine. During their participation in this study, the subjects' antibody development will be monitored.

Following vaccination with Valneva's VLA1553 vaccine, subjects may acquire immunity to CHIKV as indicated by antibody levels above a pre-defined threshold indicative of protection.

Based on the results of non-clinical studies and epidemiological data it is anticipated that a substantial number of subjects will be protected against CHIKV infection following participation in the study. However, because protection following vaccination has not yet been proven, subjects planning to travel to CHIKV endemic areas should be counseled to apply personal protective measures against mosquito bites.

An additional benefit for subjects involved in this study is derived from safety monitoring and follow-up as prophylactic measure for an early diagnosis of illness.

#### 10.5.2 Possible Benefits for Society

CHIKV is currently regarded as one of the most-likely re-emerging viruses to spread globally (Simon, Savini et al. 2008), an issue which raises an urgent demand for efficient prophylaxis. However, at present there is no treatment or vaccine available against this CHIKV-induced debilitating disease and its various symptoms (Weaver, Osorio et al. 2012; Ahola, Couderc et al. 2015; Weaver and Lecuit 2015). Thus, morbidity due to this virus is a serious threat to global health and CHIKV has now been listed as a priority pathogen by the National Institutes of Allergy and Infectious Disease (NIAID) in the United States (Ahola, Couderc et al. 2015; Weaver and Lecuit 2015; NIAID October 26, 2016). Due to

the increasing frequency and risk of CHIKV, the development of a safe and effective vaccine is a high priority.

Through their participation in this Phase 3 study, the subjects will contribute to the development of a novel vaccine against chikungunya. This Lot-to-Lot study is within a complete clinical development program, which is intended to lead to subsequent licensure of the VLA1553 vaccine, if it is shown to be safe and efficacious.

## 10.5.3 Possible Risks / Inconveniences for the Subject

VLA1553 is a live-attenuated vaccine where the attenuation of the virus leads to a reduced replication capability of the vaccine. Thus, as demonstrated in pre-clinical studies, viremia was delayed and strongly reduced and no clinical manifestations typically associated with wt CHIKV infections occurred in non-human primates. Viremia was observed in some subjects in the Phase 1 study albeit short-lived and greatly reduced from levels observed after natural infection. Only a single subject shed virus in urine.

Overall the vaccine was well-tolerated in a healthy adult population aged 18 to 45 years following a single vaccination at the low and medium dose level.

Solicited systemic reaction rates in the medium dose group were reported in 40.0% of subjects after the single vaccination. The most frequently reported symptoms of related systemic reactions (occurring at a frequency of ≥1:10) were headache, fever, fatigue and myalgia reported in 23.3%, 20.0%, 16.7% and 13.3% of subjects in the medium dose group, respectively. The majority of reactions were transient and of mild or moderate severity. For 13.3% of subjects, neutropenia, leukopenia and/or lymphocytopenia were reported as clinically relevant laboratory parameter deviations, without associated clinical signs or symptoms.

Few solicited injection site reactions (6.7%) were reported by two subjects in the medium dose group after the single vaccination. All solicited injection site reactions were of mild severity.

Allergic reactions to components of the vaccine or - in the worst case - an anaphylactic shock cannot be excluded, although such reactions have been reported in very rare cases with other vaccinations.

The possibility that vaccination may activate an autoimmune disease (e.g. multiple sclerosis) in predisposed subjects cannot be excluded.

In addition, as with any IMP, there may be unforeseeable risks associated with the use of the VLA1553 vaccine.

The blood draws performed during the study carry the possible risks of pain, hematoma, and in very rare cases an infection at the venipuncture site. The process of vaccination may also trigger syncope.

For further details on known and potential risks of this investigational product, please refer to the Investigator's Brochure.

### 10.6 COVID-19 Management

The ongoing COVID-19 pandemic may impact the conduct of this clinical study. Therefore, the study Sponsor will continuously monitor and evaluate the development of the COVID-19 pandemic in the area of the study sites.

The safety of the subject has highest priority. The study Sponsor will modify the study conduct accordingly, if any potential safety issues arise. These decisions may include halting trial recruitment or the change of subject monitoring during the study. In all cases, the subject and/or the legal representative(s) will be informed.

To protect the subject's safety, welfare, and rights, the study Sponsor will continuously evaluate specific circumstances, such as the ability to conduct appropriate safety monitoring or the potential impact on the IMP supply chain.

Depending on the local situation, subjects may not be able to come to the site for protocol-specified visits. Therefore, existing processes will be modified or new processes will be implemented. Such modifications include, but are not limited to, alternative methods of safety assessments (e.g. switching in-person visits to phone calls or virtual visits, or alternative location for assessment, including local labs) or employ mobile teams to collect serum samples. In all cases, the subject and/or the legal representative(s) will be informed.

To mitigate risks to the subjects or in response to local governmental recommendations further recruitment can be temporarily halted or some assessments will be delayed. All alternative processes will be consistent with the protocol to the extent possible.

Changes in study visit schedules, missed visits or subject discontinuations due to COVID-19 will be recorded. In addition, the reason for the implementation of any contingency measures will be documented.

Moreover, the Sponsor will communicate any measures or modifications of the study protocol to the relevant CA and IRB in line with local requirements.

The COVID-19 measures are based on the FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Public Health Emergency (as of 02-July-2020) and will be adjusted, if needed.

#### 11. STUDY PURPOSE AND OBJECTIVES

#### 11.1 Study Purpose

The purpose of the study is to demonstrate Lot-to-Lot manufacturing consistency of the final dose of the live-attenuated CHIKV vaccine candidate (VLA1553) in a healthy CHIKV-naïve population aged 18 to 45 years.

The outcome shall provide the basis for licensure of the vaccine.

## 11.2 Primary Objective

The primary objective is to demonstrate Lot-to-Lot manufacturing consistency of a live-attenuated CHIKV vaccine candidate (VLA1553) in terms of GMT 28 days following vaccination in a healthy population aged 18 to 45 years after a single immunization.

## 11.3 Secondary Objective

The secondary objective is to evaluate immunogenicity and safety of VLA1553 up to 180 days following vaccination in a healthy population aged 18 to 45 years after a single immunization.

#### 12. STUDY DESIGN

## 12.1 Overall Study Design

This is a prospective, randomized, double-blinded, multicenter Phase 3 clinical study investigating three Lots of VLA1553 at the final dose (target 1x 10E4 TCID<sub>50</sub> per 0.5 mL). Overall, approximately 402 subjects will be enrolled (i.e. ICF signed) into the study, approximately 134 subjects per VLA1553 Lot (**Table 3**).

Subjects will be block-randomized in a 1:1:1 ratio into the three study arms to receive either of three Lots of VLA1553 as a single i.m. vaccination on Day 1 (Visit 1).

All subjects will be asked to return to the study site at Day 8 (Visit 2), Day 29 (Visit 3), Day 85 (Visit 4) and Month 6 (Day 180, Visit 5) for immunogenicity sampling. Safety data collection will capture solicited AEs until Day 11 and unsolicited AEs up to Day 180 (Month 6, Visit 5) from all subjects. AESIs will be captured 2 to 21 days post-vaccination. Subjects presenting with acute arthralgia within this time period will be followed-up until resolution and monitored for recurrences until the end of the study. SAEs will also be assessed until the end of the study (Month 6, Visit 5).

Table 2 below illustrates the subject distribution scheme.

| Table 3. Subject Distribution | | | | | |
|---|---|---|---|---|---|
| Study<br>Arms | Vaccine | Cohort | Number of<br>subjects (n) | Target Dose<br>(TCID₅₀/dose) | Injection<br>Volume (mL) |
| 1 | VLA1553 | Lot 1 | 134 | - 1x 10E4 TCID₅o<br>per 0.5<br>- mL | 0.5 |
| 2 | VLA1553 | Lot 2 | 134 | | 0.5 |
| 3 | VLA1553 | Lot 3 | 134 | | 0.5 |
| | | Total N: | 402 | | |

The clinical study design is displayed in the **Figure 1** below.



Figure 1. Study Design Lot-to-Lot Consistency Study VLA1553-302

## 12.2 Study Duration

The overall duration of the study is estimated to be approximately 8 months from study initiation (first subject enrolled) to study completion (last subject last visit).

The individual subject participation is approximately 7 months from enrollment to study completion unless prematurely discontinued.

### 12.3 Study Endpoints

## 12.3.1 Primary Endpoint

### **Immunogenicity**

The primary endpoint is the Geometric mean titer (GMT) of CHIKV-specific neutralizing antibodies as determined by µPRNT assay on Day 29 post-vaccination in subjects who tested negative for CHIKV antibodies at baseline.

## 12.3.2 Secondary Endpoints

#### **Immunogenicity**

The following secondary immunogenicity endpoints will be evaluated:

- Immune response as measured by CHIKV-specific neutralizing antibody titers on Day 8, Day 85 and Month 6 post-vaccination as determined by μPRNT assay;
- Proportion of subjects with seroprotective levels (defined as baseline negative subjects) at Days 8, 29, 85 and Month 6 post-vaccination by μPRNT assay;
- Proportion of subjects with seroconversion at Day 29 and Month 6 as determined by μPRNT assay (seroconversion defined as CHIKV-specific neutralizing antibody titer of for baseline negative subjects and for baseline positive subjects);
- Fold increase of CHIKV-specific neutralizing antibody titers determined by μPRNT assay at Days 8, 29, 85 and Month 6 post-vaccination as compared to baseline;
- Proportion of subjects reaching an at least 4-fold, 8-fold, 16-fold or 64-fold increase in CHIKV-specific neutralizing antibody titer compared to baseline as measured by μPRNT assay.

#### Safety:
- > Frequency and severity of solicited injection site and systemic reactions within 10 days post-vaccination;
- > Frequency and severity of unsolicited adverse events (AEs) within 28 days post-vaccination;
- Frequency and severity of any AE during the entire study period;
- Frequency and severity of any serious adverse event (SAE) during the entire study period;
- Frequency and severity of any adverse event of special interest (AESI) within 2 to 21 days post-vaccination.

### 12.4 Randomization and Blinding

The approximately 402 subjects will be block-randomized into the three study arms in a ratio of 1:1:1 at Visit 1 as described in Section 12.1.

In order to minimize/avoid bias, assignment into one of these study arms will be blinded for these subjects and the site staff, as well as the biostatistician (i.e. double-blind).

Each subject will have a unique subject identification code obtained from the interactive voice response system/interactive web response system (IXRS) assigned at the screening visit. The Investigator will keep a record (i.e. the subject screening log) of subjects who entered screening.

Randomization will be performed via the IXRS. At Day 1 (Visit 1, day of vaccination) eligible subjects will be assigned to the respective IMP Lot.

An overview of persons who will be (un)blinded is provided below:

# Unblinded:

- > DSMB voting members;
- ➤ Bio-statistician preparing unblinded analysis for the DSMB.

# Blinded:

- ➤ Investigators and all other study staff involved in study conduct, safety assessments and IMP handling (i.e. perform preparation of the study vaccine, maintain the drug accountability logs detailing the dates and quantities of IMP administered to each subject);
- > Study participant;
- ➤ Bio-statistician (except the one involved in DSMB);
- ➤ CRA's responsible for monitoring study data, IMP handling and verifying drug accountability (during the study and performing overall drug accountability);

- ➤ All laboratory personnel at central laboratories for safety and immunogenicity laboratory assessments;
- >All other Sponsor and CRO staff including medical monitor and laboratory personnel at the Sponsor's labs for additional testing procedures.

## 12.4.1 Blinding Process

Vials are provided to the sites in a blinded manner in order to ensure the blinding of study participants, site staff performing the safety assessments and site staff performing IMP preparation and administration. Identification of the syringe is guaranteed by placing a tear-off label containing Kit number, Subject number, date of injection and operator onto the label.

For further details please refer to the IMP Manual.

## 12.4.2 Unblinding

The randomization assignment is not to be revealed except in emergency cases in which unblinding is necessary for the clinical management of an SAE. In such events, Investigator must either inform the Sponsor before breaking the blind or immediately after unblinding has been performed.

In case of emergency, the vaccine administered to the subjects can be revealed through the web-response system (IXRS).

### 12.5 Study Termination - Study Stopping Rules

The study may be paused or prematurely terminated, after consultation with the DSMB, if vaccine-related SAEs or other significant vaccine-related side effects occur. In addition, the Sponsor may stop the entire study for any reason at any time.

If the Sponsor or Investigator decides to terminate the study before it is completed, they will notify each other in writing, stating the reasons for early termination. In terminating the study, the Sponsor and the Investigator will ensure that adequate consideration is given to the protection of the subjects' interests. The Sponsor or Investigator will notify the relevant regulatory authorities or IRB in writing in accordance with local requirements. Documentation will be submitted for filing in the Investigator File and the Trial Master File.

#### 13. SUBJECT SELECTION, WITHDRAWAL AND DISCONTINUATION

Approximately 402 adults of either gender, who satisfy the inclusion and exclusion criteria listed below will be invited to participate in the study.

#### 13.1 Inclusion Criteria

Subjects who meet ALL of the following criteria are eligible for this study:

- 1. Subject is 18 to 45<sup>vi</sup> years of age on the Day of screening (Visit 0);
- Subject has an understanding of the study and its procedures, agrees to its provisions, and gives voluntarily written informed consent prior to any study-related procedures;
- 3. Subject is generally healthy<sup>vii</sup> as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests;
- 4. If subject is of childbearing potential:
  - a) Subject has practiced an adequate method of contraception (see below) during the 30 days before screening (Visit 0);
  - b) Subject has a negative serum or urine pregnancy test at screening (Visit 0) or Visit 1, respectively;
  - c) Subject agrees to employ adequate birth control measures for the first three months post-vaccination (i.e. until Day 85, Visit 4). This includes one of the following measures:
    - Hormonal contraceptives (e.g. implants, birth control pills, patches);
    - Intrauterine hormone-release systems or intrauterine device;
    - Barrier type of birth control measure (e.g. diaphragms, cervical caps);
    - Vasectomy in the male sex partner ≥ 3 months prior to first vaccination.
    - Sexual abstinence;
    - Same sex relationships;
    - Condoms when used in combination with any of the female contraceptive measures outlined above<sup>viii</sup>.

#### 13.2 Exclusion Criteria

Subjects who meet ANY of the following criteria are NOT eligible for this study:

vi From the 18th birthday until the last day before the 46th birthday.

Vii Subjects are considered *generally healthy* if (1) any chronic illness/condition, e.g. hypertension, type 2 diabetes mellitus, or hyperlipidemia is stable and well-controlled on therapy for the past 6 months, and (2) they do not have a disease that is identified as an exclusion criterion.

viii Condoms are not to be used as a sole means of contraception.

- Subject has had a CHIKV infection in the past (self-reported), including suspected CHIKV infection; is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical study involving an investigational CHIKV vaccine;
- 2. Subject has an acute or recent infection (and who is not symptom-free in the week prior to the Screening Visit (Visit 0);
- 3. Subject tests positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
- Subject has received another live virus vaccine within 28 days or inactivated vaccine within 14 days prior to vaccination in this study or plans to receive a vaccine within 28 days or 14 days after vaccination, respectively;
- Subject has abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the study based on his/her judgement;
- 6. Subject has a medical history of or currently has acute or progressive, unstable or uncontrolled clinical conditions (e.g. cardiovascular, respiratory, neurologic, psychiatric, or rheumatologic conditions) that poses a risk for participation in the study, based on Investigators clinical judgement. Examples include individuals with poorly controlled or unstable disease, ongoing suspected or active inflammation, or poor compliance with pharmacologic treatment, or presence of high risk comorbidities (e.g. significant cardiopulmonary disease);
- 7. Subject has a history of immune-mediated or clinically relevant arthritis/arthralgia:
- 8. Subject has a history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the subject may be enrolled. A history of hematologic malignancy is a permanent exclusion. Subjects with a history of skin cancer must not be vaccinated at the previous tumor site;
- 9. Subject has a known or suspected defect of the immune system, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day within 4 weeks prior to study entry, radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous 3 years; topical and inhaled steroids are allowed.

- Subject has a history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications);
- 11. Subject presents with clinical conditions representing a contraindication to intramuscular vaccination and blood draws;
- 12. Subject is pregnant (positive serum or urine pregnancy test at screening or Visit 1, respectively), has plans to become pregnant during the first three months post-vaccination or lactating at the time of enrollment;
- 13. Subject has donated blood, blood fractions or plasma within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or plans to donate blood or use blood products until Day 180 of the study;
- 14. Subject has a rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating;
- 15. Subject has a known or suspected problem with alcohol or drug abuse as determined by the Investigator;
- 16. Subject has any condition that, in the opinion of the Investigator, may compromise the subjects well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
- 17. Subject is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
- 18. Subject has participated in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study;
- 19. Subject is a member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

### 13.3 Delay Criteria for Vaccination

Vaccination will be delayed if:

 Subject has an acute febrile infection within 72 hours prior to vaccination or oral temperature greater than or equal 38.0 °C/ 100.4 °F on the day of vaccination (subject may be rescheduled within the screening visit window until subject has completed 72 hours of no fever);

- 2. Subject has received antipyretics within 4 hours prior to the scheduled time of vaccination (subject may be rescheduled within the screening visit window).
- 3. Subject has received any live or inactivated vaccine within 28 days or 14 days prior to vaccination, respectively.

In addition, for a rescheduled vaccination all inclusion and none of the exclusion criteria must be met; in case not all of these criteria are met, the subject will be excluded from the study.

The rescheduled visit should be within the specified time window for the vaccination visit. In case the time window for the rescheduled visit cannot be met, the subject might be invited for a re-screening.

Subjects who have been screen failed under protocol version 2.0 due to the site not receiving the subjects CHIKV-serostatus from the testing laboratory within the 28 day screening window can be asked back for re-screening. All eligibility tests will again be performed with the exception of the CHIKV-serostatus test<sup>ix</sup>

Moreover, re-screening will not be allowed for subjects who screen fail due to other reasons, such as inclusion/exclusion criteria.

## 13.4 Pregnancy Testing and Birth Control

The risk of maternal-to-fetal transmission of chikungunya vaccine virus during pregnancy cannot be excluded. Therefore, only women of childbearing potential presenting with a negative pregnancy test and practicing the use of adequate birth control before conduct and during the first three months of the study are eligible for inclusion into the study.

A woman is considered of childbearing potential if fertile, following menarche and until becoming post-menopausal unless permanently sterile.

Women of childbearing potential must have practiced an adequate contraceptive method during the 30 days before Visit 0 (Screening Visit) and the first three months until Visit 4 (Day 85/ Month 3) and present with a negative **serum** pregnancy test at Visit 0 (Screening Visit), a negative **urine** pregnancy test prior to vaccination. In addition, a **urine** pregnancy test will need to be performed at the Early Termination Visit (if applicable).

Women of childbearing potential are required to practice an acceptable method of birth control for the first three months post-vaccination. An acceptable method of birth control is defined as those, which result in a low failure rate when used consistently and correctly.

This includes one of the following measures:

<sup>ix</sup> The original CHIKV result from the sample taken at the initial screening visit will be valid for up to 60 days from sample collection.

Valneva Austria GmbH

CONFIDENTIAL

- > Hormonal contraceptives (e.g. implants, birth control pills, patches);
- Intrauterine hormone-releasing system or intrauterine device;
- > Barrier type of birth control measure (e.g. diaphragms, cervical caps);
- ➤ Vasectomy in the male sex partner ≥ 3 months prior to first vaccination;
- Sexual abstinence:
- Same-sex relationships.
- Condoms when used in combination with any of the female contraceptive measures outlined abovex.

Women without childbearing potential are not required to perform any birth control measure. A woman is considered of non-childbearing potential, if she is:

- Surgically sterilized for ≥ 3 months prior to Visit 1 (permanent sterilization methods include hysterectomy, bilateral salpingectomy or bilateral oophorectomy, or transcervical sterilization (Essure and Adiana procedures), or tubal ligation;
- Postmenopausal for ≥ 1 year prior to study start as historically confirmed by a gynecologist or general practitioner.

If a subject becomes pregnant during the study, she must immediately inform the Investigator and the subject is asked to attend all remaining visits according to schedule.

# 13.5 Subject Withdrawal or Discontinuation

Any subject has the right to withdraw from the study at any time for any reason, without the need to justify. The Investigator and Sponsor also have the right to prematurely terminate a subject's further participation in the study, e. g. in the case of non-compliance or if – in the judgment of the Investigator and/or Sponsor – continued participation would pose an unacceptable risk for the subject.

The primary reason for withdrawal / discontinuation of a subject from treatment and/or from the study should be documented in the electronic Case Report Form (eCRF) (e.g. withdrawal of consent, Investigator/Sponsor recommended withdrawal, lost to follow up, death).

The primary reasons for discontinuation will be reported on the Discontinuation eCRF, including:

- ➤ Withdrawal of consent (not due to AE);
- ➤ Withdrawal due to AE:
- ➤ Lost to follow-up (defined as 3 documented unsuccessful attempts to contact the subject xi);

x Condoms are not to be used as a sole means of contraception.

- ➤ Investigator decision (e.g. non-compliance with protocol);
- > Study terminated by Sponsor;
- ➤ Death;
- > Or other (reason to be specified by the Investigator, e.g. technical problems).

Regardless of the reason, all data available for the subject up to the time of completion/discontinuation should be recorded on the appropriate CRF.

Data collected on withdrawn subjects will be used in the analysis and included in the clinical study report.

Subjects who do not complete the entire study due to withdrawal or discontinuation for any reason will not be replaced.

Valneva Austria GmbH

Note that a subject who is lost to follow-up but later returns to the study site for a follow-up can still complete the study provided he/she has received the vaccination according to the protocol.

### 14. INVESTIGATIONAL MEDICINAL PRODUCT

## 14.1 Description of VLA1553

The CHIKV vaccine (VLA1553) is a live-attenuated vaccine comprising a large deletion of 60 amino acids in the nsP3 gene encoding the non-structural replicase complex protein nsP3, which leads to attenuation of the virus *in vivo*.

VLA1553 is present in a freeze dried presentation and must be reconstituted with a solvent consisting of sterile water for injection in a prefilled syringe before use.

One dose (0.5 mL) of the VLA1553 vaccine contains between 1.6 x10E3 and 2.5 x10E4  $TCID_{50}$  per dose. The active ingredient is suspended in a formulation buffer of pH 7.3, before freeze drying.

| Table 14.1-1 Composition of the VLA1553 lyophilized Drug Product | |
|---|---|
| Active substance | |
| Live-attenuated CHIKV | Target TCID <sub>50</sub> /dose |
| Live-atteridated of fire | 1 x 10E4TCID <sub>50</sub> |
| Excipients and buffer components | Freeze Dried Formulation/ dose |
| di-Potassium Hydrogen Phosphate | 0.313 mg |
| Potassium di-Hydrogen Phosphate | 0.098 mg |
| Trisodium citrate dihydrate | 3.68 mg |
| Sucrose | 25 mg |
| Magnesium Chloride hexahydrate | 0.51 mg |
| D-Sorbitol | 2.5 mg |
| L-Methionine | 0.75 mg |
| Recombinant Human Albumin | 0.01% (equals 0.05 mg) |
| pH | 7.3 |

# 14.2 IMP Packaging, Labeling, and Storage

#### 14.2.1 VLA1553 Packaging

VLA1553 will be provided in kit containing one single-use 2R vial with the lyophilized powder of VLA1553 vaccine, one solvent consisting of 0.5 mL sterile water for injection in a prefilled syringe and a sterile needle set (i.e. 2x 25G x 1½, 0.50x40 mm) for reconstitution and administration.

### 14.2.2 IMP Labeling

VLA1553 will be labeled according to the valid regulatory requirements for clinical trials and appropriate retest dates will be assigned (MM/YYYY).

### 14.2.3 IMP Storage

VLA1553 has an expected retest date of 24 months from the date of manufacture, considering the specified storage conditions of +2-8 °C (35.6 °F to + 46.4 °F). A stability program is currently ongoing and if any impact on the stability profile are observed, the study sites will be informed accordingly. The vaccine must not be used after the retest date indicated on the package.

VLA1553 must be stored at +2-8 °C (35.6 °F to + 46.4 °F) in a refrigerator in a room not accessible to unauthorized persons. Storage at room temperature or higher should be avoided because of potential impairment to immunogenicity and tolerability. Temperature monitoring systems will be used.

## 14.2.4 Dispensing and Accountability of IMP

Current drug accountability logs have to be maintained, detailing the dates and quantities of IMP administered to each subject. Records will be maintained that include subject identification code (SIC), dispensation date, and amount dispensed. This documentation will be available to the CRA to verify drug accountability during the study and to perform overall drug accountability.

Used and unused IMP will be accounted for and returned to the CMO/Sponsor. In addition, used IMP can be destroyed on-site upon Sponsor approval.

A study specific IMP manual with further details on IMP handling will be provided.

#### 15. STUDY PROCEDURES

#### 15.1 Informed Consent and Enrollment

Any healthy volunteer who provides informed consent (i.e., signs and dates the informed consent form) is considered enrolled in the study.

The Investigator will inform the subject about the procedures, risks and benefits of the study. Fully informed, written consent must be obtained from each subject prior to any assessment being performed. It is important that the subject is allowed sufficient time to decide on his / her participation in the study.

### 15.2 Subject Identification Code

At Visit 0, a 13-character subject identification code will be assigned to each subject. The first four digits are the product identifier (e.g. 1553 for this product) provided by the Sponsor. The fifth digit indicates this study being the second Phase 3 study (e.g.1553-2), the sixth and seventh digits are site identification number (i.e. 1553-2-01). The last three digits are assigned in ascending order as the subjects are enrolled (i.e., signing the informed consent form, e.g. 1553-2-01-001).

#### 15.3 Investigational Treatment

### 15.3.1 Description of Treatment

All subjects will receive a single intramuscular vaccination in the deltoid region of the arm of VLA1553 vaccine according to the vaccination schedule as described in 24.2-1 of Study Procedures. Subjects will be assigned in a 1:1:1 ratio to one of the three study arms and will receive one of the three Lots of the final target dose level of 1 x 10E4 TCID<sub>50</sub> per 0.5 mL dose. All subjects will be followed up for approximately 6 months following the single study vaccination (see also Section 12.1).

### 15.3.2 Vaccine Preparation and Administration

VLA1553 is available as a suspension after reconstitution of targeted 1x 10E4TCID<sub>50</sub> per 0.5 mL dose.

IMP preparation and administration will be done according to the following procedure:

1. CAUTION: Preservatives, antiseptics, detergents, and other anti-viral substances may inactivate the vaccine. Use only provided sterile syringes that are free of preservatives, antiseptics, detergents, and other anti-viral substances for reconstitution and injection of VLA1553.

- 2. Before reconstitution, the lyophilized VLA1553 is a white to pale yellow compact crystalline plug. VLA1553 when reconstituted, is a clear pale to slightly yellow liquid solution.
- 3. The solvent is sterile water for injection and supplied in a 1.5 mL prefilled syringe, filled with 0.5 mL and closed with a temper evident closure system (Vetter V-OVS®) to safeguard the product integrity.
- 4. VLA1553 must be reconstituted by adding the entire content of the prefilled syringe of the solvent into the vial containing the lyophilized powder.
- 5. Twist the white temper evident closure system on the syringe bottom and remove the part of the closure system. For reconstitution, immediately attach the first provided needle on the luer lock of the syringe by twisting the needle clockwise until it locks.
- 6. Puncture the stopper of the vial with the needle on the syringe and add the entire amount of the solvent of the syringe into the vial containing the powder cake. Gently agitate the vial to dissolve completely and wait for at least one minute for complete reconstitution of the vaccine. Avoid strong shaking or vortexing. Inspect the liquid solution by visual control for any particulate matter and discoloration prior to administration.
- 7. Withdraw the entire amount from the vial of the reconstituted vaccine into the same syringe with the same attached needle.
- 8. To administer the vaccine, the second provided needle must be used. Change the needle and inject the reconstituted vaccine intramuscularly (i.m.) into the deltoid muscle as soon as possible within an allowable time window of maximal 2 hours.
- The used vials should be kept within the empty kits for drug accountability purposes. Used syringes and needles should be disposed in accordance with local requirements.

Under no circumstances should the VLA1553 vaccine be administered intravascularly, as this could lead to hypersensitivity reactions such as shock.

Anaphylaxis or other possible severe acute, post-vaccination adverse reactions to vaccines, including VLA1553 vaccine, are very rare, but can occur. Therefore, appropriate emergency equipment and medication as well as adequately trained personnel must be on site whenever a vaccination is performed.

A study specific IMP manual with further details on IMP handling will be provided.

#### 15.3.3 Post- Vaccination Observation

Following vaccination, the subject will be observed for at least 30 minutes at the study site in order to provide appropriate emergency treatment should this be necessary. In addition, vital signs including pulse rate and blood pressure while seated and at rest will be measured prior to discharge (for further information see Section 17.5). Any injection site and systemic reactions will be recorded.

Prior to leaving the study site, the subject will be instructed on the use of the respective electronic Subject Questionnaire for documentation of AEs (for further information see Section 17.3), a digital thermometer for measuring oral body temperature and a measuring device for assessing injection site reactions (at the vaccination visit only).

### 15.4 Screening and Study Visits

The overall study design is illustrated in Figure 24.1-1 (in Section 24.1). For a tabular outline of study procedures and assessments required at each visit, please see Table 15.4-1, Table 15.4-2 and Table 15.4-3 as well as the Schedule of Study Procedures and Assessments in Section 24.2.

#### 15.4.1 Part A

| Table 15.4-1 | | |
|---|---|---|
| Study VLA1553-302 Study Visit Schedule – Part A | | |
| VISIT | TIME | ACTION |
| Visit 0<br>Screening | Day -28 to 0<br>(prior to<br>Visit 1) | <ol> <li>Informed consent a</li> <li>Inclusion and exclusion criteria (Section 13.1 and 13.2)</li> <li>Demographics b</li> <li>Medical history including vaccination history c (Section 17.4.1)</li> <li>Prior and concomitant Medications (Section 17.4.2)</li> <li>Physical examination, Hand Stiffness Test d and Vital Signs c (Section 17.6 and 17.5)</li> <li>Blood draw and urine sample for: <ul> <li>Serum Pregnancy test f</li> <li>CHIK Screening c</li> <li>Safety Sample h</li> <li>HIV / HBsAg / HCV testing f</li> </ul> </li> </ol> |
| Visit 1 <sup>j</sup> | Day 1 | 1. Inclusion, exclusion and delay criteria (review) (Section 13.1, 13.2 and 13.3) 2. Medical History incl. vaccination history of (update) (Section 17.4.1) 3. Concomitant Medications (Section 17.4.2) 4. Symptom-driven physical examination, Hand Stiffness Test dand Vital Signs of (Section 17.6 and 17.5) 5. Blood draw and urine sample for: a) Urine Pregnancy test of b) Baseline Sample of color immunogenicity of limmunogenicity |

| | | Table 15.4-1 |
|---|---|---|
| | s | tudy VLA1553-302 Study Visit Schedule – Part A |
| VISIT | TIME | ACTION |
| | | 8. Post-vaccination observation (Section 15.3.3) 9. AE documentation (Section 17.2) 10. Instruct on Subject eDiary <sup>m</sup> (Section 17.3) |
| Visit 2 | Day 8<br>(+/- 1d) | <ol> <li>Review Subject eDiary (Section 17.3)</li> <li>AE documentation (Section 17.2)</li> <li>Concomitant medications (17.4.2)</li> <li>Symptom-driven physical examination and Hand Stiffness Test <sup>d</sup> (Section 17.6)</li> <li>Blood draw and urine sample for: <ul> <li>a) Immunogenicity <sup>k</sup></li> <li>b) Viremia <sup>l</sup></li> <li>c) Safety Sample <sup>h</sup></li> </ul> </li> <li>Instruct on eMemory Aid (Section 17.3)</li> </ol> |
| Visit 3 | Day 29<br>Month 1<br>(+/- 4d) | Review eDiary and eMemory Aid (Section 17.3) AE documentation (Section 17.2) Concomitant Medications (Section 17.4.2) Symptom-driven physical examination and Hand Stiffness Test <sup>d</sup> (Section 17.6) Blood draw and urine sample for: |

- Occurs at enrollment (before Screening).
- b Demographics data include year of birth, age, height, weight, BMI, gender, race and ethnicity.
- Prior vaccination against relevant traveler diseases should be documented in the Medical History, i.e. YF and JEV.
- At the screening visit, a physical examination will be performed on the following body systems being described as normal or abnormal: general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological. At subsequent visits, a symptom-driven physical examination will be performed, i.e. only in case symptom is reported by the subject, a symptom-based assessment of the affected body system(s) will be performed. A Hand Stiffness and mobility examination will be performed at all study visits irrespective of prior symptoms.
- Vital signs will include systolic and diastolic blood pressure and pulse rate while seated and at rest, and body temperature measured orally before vaccination. In addition, after an observation period of 30 minutes following vaccination pulse rate as well as blood pressure while seated and at rest will again be assessed.
- A **serum** pregnancy test will be performed for all female subjects of childbearing potential at the screening visit only and a **urine** pregnancy test will be done prior to vaccination at Visit 1 and at indicated visits [blood: 3.0 mL].
- <sup>9</sup> A CHIKV Screening Sample (5.0 mL) will be obtained at Visit 0 (Screening Visit) for CHIKV-specific ELISA testing for baseline serostatus.
- h Safety laboratory sample for standard safety laboratory assessments according to Section 17.7.1.
- A positive HIV test obtained by ELISA will have to be confirmed by a second method (e.g. Western blot or PCR).
- A Baseline Sample will be drawn for retrospective investigation of potential pre-existing antibodies including but not limited to other alphaviruses (i.e. Mayaro) or Dengue and ZIKA.
- Immunogenicity sample for CHIKV-specific neutralizing antibody titer evaluation, development of further assays or retrospective safety analysis. For further information on the preparation, storage and shipment of blood samples please refer to the instructions in the respective Laboratory Manual provided in the Investigator File.
- I Viremia plasma sample for clinically indicated retrospective investigation of viremia by RT-qPCR.
- Distribute thermometer and measuring device: Instruct subject how and when to complete the eDiary. Subject will also be instructed to immediately inform the site in case of any severe solicited AEs or other severe symptoms.
- <sup>n</sup> A COVID-19 Sample for retrospective serological Sars-CoV-2 specific antibody testing.

#### 15.4.2 Part B

| Table 15.4-2<br>Study VLA1553-302 Study Visit Schedule – Part B | | |
|---|---|---|
| VISIT | TIME | ACTION |
| Visit 4 Mont | Day 85<br>Month 3<br>(+/- 7d) | <ol> <li>Review eMemory Aid (Section 17.3)</li> <li>AE documentation (Section 17.2)</li> <li>Concomitant Medications (Section 17.4.2)</li> <li>Symptom-driven physical examination and Hand Stiffness Test (Section 17.6)</li> <li>Blood draw for and urine sample for: <ul> <li>a) Urine Pregnancy test <sup>a</sup></li> <li>b) Immunogenicity <sup>b</sup></li> <li>c) Safety Sample <sup>c</sup></li> </ul> </li> </ol> |
| Visit 5 | Day 180<br>Month 6<br>(+/- 14d) | <ol> <li>Review eMemory Aid (Section 17.3)</li> <li>AE documentation (Section 17.2)</li> <li>Concomitants Medication (Section 17.4.2)</li> <li>Symptom-driven physical examination and Hand Stiffness Test (Section 17.6)</li> <li>Blood draw and urine sample for: <ul> <li>a) Urine Pregnancy test <sup>a</sup></li> <li>b) Immunogenicity <sup>b</sup></li> <li>c) Safety Sample <sup>c</sup></li> <li>d) COVID-19 Sample <sup>d</sup></li> </ul> </li> </ol> |

- <sup>a</sup> A **urine** pregnancy test will be performed for all female subjects of childbearing potential at indicated visits.
- Immunogenicity sample for CHIKV-specific neutralizing antibody titer evaluation, development of further assays or retrospective safety analysis. For further information on the preparation, storage and shipment of blood samples please refer to the instructions in the respective Laboratory Manual provided in the Investigator File.
- Safety laboratory sample for standard safety laboratory assessments according to Section 17.7.1.
- d A COVID-19 Sample for retrospective serological Sars-CoV-2 specific antibody testing.

#### 15.4.3 Unscheduled Visit

An unscheduled visit can be held at any time during the study if deemed necessary by the Investigator (e.g. follow-up on unexpected AEs or SAEs) or the DSMB. Assessments performed at an unscheduled visit will be at the Investigator's or DSMB's discretion. Unscheduled visits and any procedures/assessments performed during such a visit (e.g. physical examination, laboratory test) should be documented in the source data and the eCRF.

## 15.4.4 Early Termination Visit

Subjects who terminate participation or who are withdrawn from the study prematurely will undergo investigations as outlined below during an Early Termination Visit, if possible. Every effort should be made to have discontinued subjects complete the study Early Termination (ET) Visit (see Table 15.4-3).

| Table 15.4-3 Study VLA1553-302 Study Visit Schedule – Early Termination | | |
|---|---|---|
| VISIT | TIME | ACTION |
| ET | nnscheduled | <ol> <li>Review Subject eDiary or eMemory Aid, as applicable (Section 17.3)</li> <li>AE/AESI/SAE documentation (Section 17.2)</li> <li>Concomitant Medications (Section 17.4.2)</li> <li>Symptom-driven physical examination and Hand Stiffness Test (Section 17.6)</li> <li>Blood draw and urine sample for: <ul> <li>a) Urine Pregnancy test <sup>a</sup></li> <li>b) Immunogenicity <sup>b</sup></li> <li>c) Viremia <sup>c</sup></li> <li>d) Safety Sample <sup>d</sup></li> <li>e) COVID-19 Sample <sup>e</sup></li> </ul> </li> <li>Documentation of reason for early termination</li> </ol> |

- <sup>a</sup> A urine pregnancy test will be performed for all female subjects of childbearing potential at indicated visits.
- b Immunogenicity sample] for CHIKV-specific neutralizing antibody titer evaluation, development of further assays or retrospective safety analysis. For further information on the preparation, storage and shipment of blood samples please refer to the instructions in the respective Laboratory Manual provided in the Investigator File.
- Only if the ET visit occurs prior to Day 29, a viremia plasma sample should be obtained from the subject for clinically indicated retrospective investigation of viremia by RT-qPCR.
- Safety laboratory sample for standard safety laboratory assessments according to Section 17.7.1
   A COVID-19 Sample for retrospective serological Sars-CoV-2 specific antibody testing.

In case an ET Visit is not possible, a follow-up safety phone call should be made as soon as possible after termination to capture at least concomitant medications and solicited and unsolicited AEs since the last study visit.

The reason for early termination should be clarified in as much detail as possible. If an AE was the reason for early study termination details on that specific AE(s) should be captured (see Section 13.5). The reason for discontinuation will be recorded on the eCRF, and data collected up to the time of discontinuation will be used in the analysis and included in the clinical study report.

In the event of subject discontinuation due to an AE, clinical and/or laboratory investigations that are beyond the scope of the required study observations/assessments may be performed as part of the evaluation of the event. These investigations will take place under the direction of the Investigator in consultation with the Sponsor, and the details of the outcome may be reported to the appropriate regulatory authorities by the Sponsor.

### 15.5 Procedures for Monitoring Subject Compliance

All study procedures are to be performed under the supervision of the Investigator at the study site, and thus, no separate procedures will be used to monitor subject compliance.

#### 16. ASSESSMENT OF IMMUNOGENICITY

All serum samples for neutralization titer determination will be handled according to the procedures supplied to each investigative site for the preparation, storage and shipment of samples (refer to Laboratory Manual). Each clinical study site will be responsible for the separation of serum from whole blood samples and the safe and controlled storage of serum samples prior to shipment to the central analytical laboratory.

At the end of the study, results of immunogenicity assessments will be provided to the Investigator.

Immunogenicity assessment measuring neutralizing antibodies will be performed on samples collected at Days 1, 8, 29 (Month 1), 85 (Month 3) and 180 (Month 6) after a single immunization.

#### 16.1 Determination of vaccine-induced neutralizing antibody response

Immunogenicity of VLA1553 will be evaluated using a micro Plaque Reduction Neutralization Test (μPRNT), which is based on the same principle as a plaque reduction neutralization assay (PRNT), but allows testing with higher throughput. This assay differs from the μNT assay used for the assessment of neutralizing antibodies during Phase 1 clinical testing. Chikungunya virus neutralizing antibodies will be measured in the μPRNT using a serially passaged, live-attenuated CHIKV vaccine (CHIKV 181/25, TSI-GSD-218 or 181/clone 25) developed by the Walter Reed Army Institute of Research (WRAIR, US).

The CHIKV µPRNT evaluates the levels of antibodies that neutralize CHIKV infection of Vero cells in human serum samples.

Seven (7) two-fold serial dilutions of the de-complemented serum samples are prepared in round-bottom 96-well plates. CHIKV 181/25 at a target working dilution (to obtain 100 PFU/well) is added sequentially to the serum dilutions and incubated at 37°C and 5% CO<sub>2</sub> for 60 minutes. Serum-virus complexes are then transferred onto plates, previously seeded overnight with Vero cells, and incubated at 37°C and 5% CO<sub>2</sub> for 60 minutes. Then, the serum-virus complexes are removed and a virus maintenance medium containing 0.5% Methyl Cellulose is added to the wells, followed by an incubation of 17 ± 1 hours at 37°C and 5% CO<sub>2</sub>. The following day, cells are fixed with 4% Paraformaldehyde for 15 minutes and permeabilized with 0.2% Triton X-100. Following cell permeabilization, indirect immunostaining is performed. Primary antibody diluted in blocking agent is added to the plates and incubated at 37°C for 60 minutes. Afterwards, the secondary antibody diluted in blocking agent is added to the plates and incubated at 37°C for 30 minutes. Substrate is

added to the plates and incubated for 10 minutes in the dark. Plates are rinsed with sterile water and left to be dried completely. Images from each well are acquired by an automated microscope system (ScanLab reader). The number of resulting PFUs in the wells is inversely proportional to the level of functional antibodies present in the serum, which is directly proportional to the immunological response of the subject.

The cut-off of CHIKV-specific neutralization antibody titer to be used in the analysis of seroconversion is defined as CHIKV-specific neutralizing antibody titer of baseline negative subjects. Seroconversion for baseline positive subjects is defined as a increase over baseline.

### 16.2 Additional Testing Procedures

Serum samples obtained in this study may, in addition to its use for assessment of CHIKV-specific neutralizing antibody titers, also be used for further development of the vaccine, including but not limited to the following assays:

- Passive immunization assays to evaluate the potency of immune sera to protect animals from infection after wild-type challenge;
- Development of additional neutralization assays (e.g. μNT, PRNT, virus replicon particle neutralization assays) for the assessment of cross neutralization of heterologous CHIKV strains or other related (alpha) viruses;
- Detection of anti-CHIKV antibodies by enzyme linked immunosorbent assay (ELISA);
- Detection of viremia by viral culture;
- CHIKV sequencing;
- Clinical diagnostic work-up.

Such development may occur at laboratories other than the central analytical laboratory used for this study.

#### 17. ASSESSMENT OF SAFETY

#### 17.1 Definitions

#### 17.1.1 Adverse Events

An adverse event (AE) is defined as any untoward medical occurrence in a subject administered an investigational product that does not necessarily have a causal relationship with the treatment. All new abnormalities or any exacerbation in intensity or frequency (worsening) of a pre-existing condition during or after vaccination have to be documented as AEs.

#### 17.1.2 Serious Adverse Event

A **serious** adverse event (SAE) is defined as any untoward medical occurrence that at any dose meets one or more of the following criteria:

- Outcome is fatal/results in death (including fetal death);
- Is life-threatening defined as an event in which the subject was, in the judgment of the Investigator, at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death had it been more severe:
- Requires inpatient hospitalization or results in prolongation of an existing hospitalization;
- Results in persistent or significant disability/incapacity (i.e., a substantial disruption of a person's ability to conduct normal life functions);
- Results in congenital anomaly/birth defect;
- Is a medically important condition a medical event that may not be immediately life-threatening or result in death or require hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the definitions above. This definition also applies to progression of disease leading to a serious outcome.

In case of hospitalization or prolonged hospitalization for diagnostic or elective medical procedures that were planned prior to vaccination to treat a pre-existing condition that did not change in severity, neither the condition leading to the hospitalization or prolonged hospitalization, nor the medical procedure itself need to be reported as an SAE. In this case, the underlying diagnosis or condition should be reported in the medical history section of the eCRF and the corresponding medical procedure should be documented as a comment to the underlying diagnosis or condition in the eCRF's medical history section.

The Sponsor will classify the SAEs as either expected or unexpected:

➤ Expected: An AE that is listed in the current Investigator's Brochure (IB);

➤ Unexpected: An AE that is not listed in the current IB, or it differs because of

greater severity or greater specificity.

For the purpose of this study, AEs graded as potentially life-threatening (Grade 4) (see Section 17.2.2 for solicited AEs) will be reported as SAEs.

### 17.1.3 Adverse Events of Special Interest

An AESI (serious or non-serious) is an event of scientific and medical concern specific to the Sponsor's product.

### 17.1.4 Medically-Attended Adverse Event

All AEs where subjects are seeking medical care (i.e. doctor's office, emergency service, hospital, but not including use of self-medication).

## 17.1.5 Preexisting Diseases

Preexisting diseases that are present before entry in to the study, that are described in the medical history, and that manifest with the same severity, frequency, or duration after vaccine exposure, will not be recorded as AEs. Furthermore, routine health checks required due to pre-existing diseases will not be recorded. However, when there is an increase in the severity of a preexisting disease, the event must be described on the AE CRF page.

### 17.1.6 Untoward Medical Occurrences Not Considered Adverse Events

Each untoward medical occurrence experienced <u>before</u> vaccine exposure (for example, from the time of signed informed consent up to but not including vaccine exposure) will be described in the medical history.

#### 17.2 Collection, Documentation and Assessment of Adverse Events

#### 17.2.1 Unsolicited Adverse Events

Subjects will be provided with an eDiary and eMemory Aid to collect unsolicited AEs occurring until the end of study (Visit 5, see Section 17.3). Additionally, the Investigator will enquire about AEs during study visits. Clinically relevant laboratory parameter changes constitute unsolicited AEs, too, unless they are considered a symptom of an underlying AE or part of a syndrome that is reported as AE (e.g. presence of blood cells in urine in a

person diagnosed with urinary tract infection). In addition, symptoms noted during the symptom-driven physical exams (unless already covered by an AE) constitute AEs.

All unsolicited AEs need to be documented in the respective AE section of the eCRF during applicable study visit (Visits 1 to 5 or unscheduled visit(s), if applicable), regardless of their source (AEs noted in the eMemory Aid (see Section 17.3), open question to subject, laboratory parameters, symptom-driven physical examination).

Any symptom is regarded as a separate AE. However, if the Investigator considers several symptoms to be in the context of one underlying diagnosis, the Investigator may merge these symptoms into one single appropriate AE. The AE term entered into the eCRF should contain all symptoms summarized to one event (e.g. "Influenza with flu-like-symptoms, fever and headache").

The Investigator will follow-up on each AE until it is resolved or until the medical condition of the subject is stable. All relevant follow-up information will be reported to the Sponsor until the end of the study for each subject. SAEs ongoing at the time of Visit 6 will be followed until resolution or achievement of stable clinical conditions, latest until the end of the study.

Beyond study end, if the investigator becomes aware of SAEs that are fatal, life-threatening or suspected to be related to study treatment will continue to be reported until 6 months after the last study visit of the respective subject (i.e., Visit 5).

The following information will be documented for each AE: severity, causality, outcome, seriousness, medically-attended, action taken to treat AE, start and stop dates.

#### 17.2.1.1 Severity

The investigator will assess the severity of AEs using his/her clinical expertise and judgment based on the most appropriate description below:

Mild (Grade 1): Awareness of signs or symptoms, but easily tolerated, does not

interfere with daily activities.

Moderate (Grade 2): Discomfort enough to interfere with usual activity and with or

without requiring medical intervention.

Severe (Grade 3): Incapable of work or usual activity and requiring medical

intervention.

### 17.2.1.2 Causality

Causality is a determination of whether there is a reasonable possibility that the vaccine administration is etiologically related to/associated with the AE.

For AEs, the Investigator will assess the causal relationship between the IMP and the AE using his/her clinical expertise and judgement according to the following most appropriate algorithm for the circumstances of the AE:

Probable: Reaction that follows a reasonable temporal sequence from

administration of the IMP, or that follows a known or expected response pattern to the suspected treatment and that could not reasonably be explained by known characteristics of the

subject's clinical state.

Possible: Reaction that follows a reasonable temporal sequence from

administration of the IMP, or that follows a known or expected response pattern to the suspected treatment; but that could

readily have been produced by a number of other factors.

Unlikely: Reports not following a reasonable temporal sequence from

administration of the IMP; an event, which may have been

produced by the subject's clinical state or by other

environmental factors. A more likely alternative etiology exists.

Not related (unrelated): Events for which sufficient information exists to conclude that the

etiology is unrelated to the IMP.

An alternative aetiology, especially COVID-19 related symptoms, should be taken into consideration for a thorough causality assessment by the Investigator. Current symptoms include fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea. For latest case definitions please refer to CDC webpage (https://www.cdc.gov/coronavirus/2019-ncov/symptoms-testing/symptoms.html). These symptoms need to be documented in the eCRF.

AEs with a causality reported as probable or possible will be considered related to the IMP. AEs with missing causality assessment will be regarded as related unless further specified. All other AEs will be considered as not related to IMP.

#### 17.2.1.3 Assessment and Outcome of Adverse Events

Each AE from vaccination until study completion/termination will be described on the AE eCRF (i.e., 1 AE per form) using the medical diagnosis (preferred), symptom, or sign, in standard medical terminology in order to avoid the use of vague, ambiguous, or colloquial expressions (see definition in Section 17.1.1). AEs will be evaluated by the Investigator for:

- > Seriousness as defined in Section 17.1.2
- > Severity as defined in Section 17.2.1.1
- Causal relationship to vaccine exposure as defined in Section 17.2.1.2

For each AE, the outcome will also be documented as either:

> recovering/resolving

> recovered/resolved

> recovered/resolved with sequelae

> not recovered/not resolved

> fatal

> unknown

If the severity rating for an ongoing AE changes before the event resolves, the AE will not be reported a second time. Instead the original AE entry will be revised. For purposes of data capture the highest severity rating during the course of a single AE will be the severity rating entered on the AE eCRF.

**NOTE:** A subject's death per se is not an event, but an outcome. The event which resulted in the subject's death must be fully documented and reported, regardless of being considered related to treatment or not.

#### 17.2.2 Solicited Adverse Events

### 17.2.2.1 Injection Site Reaction – Measurement and Evaluation

Subjects will be provided with a measuring device to measure the size of any measurable injection site reaction that may develop after vaccination. The subject will be instructed on how to measure any such reactions over a period of 10 consecutive days starting on the day of vaccination along the longest diameter of the reaction area and record this measurement in the Subject eDiary. Injection site reactions include injection site pain, tendemess, erythema/redness, induration and swelling.

Injection site reactions will be rated based on the FDA Guidance on Toxicity Grading Scales as described in Table 17.2-1. Any grade 4 injection site reaction should be reported as an SAE (see Section 17.1.2).

Table 17.2-1
Grading of Injection Site Reactions – Vaccine Specific Criteria

| Ordania of injection ofte reactions – vaccine opecine oftena | | | | |
|---|---|---|---|---|
| Vaccine-specific<br>Criteria | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening<br>(Grade 4)° |
| Pain | Does not interfere with activity | Repeated use of<br>non-narcotic pain<br>reliever > 24 hours<br>or interferes with<br>activity | Any use of narcotic pain reliever or prevents daily activity | Emergency room<br>(ER) visit or<br>hospitalization |
| Tenderness | Mild discomfort to touch | Discomfort with movement | Significant<br>discomfort at rest | ER visit or hospitalization |
| Erythema /<br>Redness <sup>a</sup> | 2.5 – 5.0 cm<br>0.98 – 1.96 inch | 5.1 – 10.0 cm<br>1.97 – 3.94 inch | > 10.0 cm<br>> 3.94 inch | Necrosis or exfoliative dermatitis |
| Induration /<br>Swelling <sup>b</sup> | 2.5 – 5.0 cm<br>(0.98–1.96 inch)<br>and does not<br>interfere with<br>activity | 5.1– 10.0 cm<br>(1.97 – 3.94 inch)<br>or interferes with<br>activity | > 10.0 cm<br>(> 3.94 inch) or<br>prevents daily<br>activity | Necrosis |

a In addition to grading the measured local reactions at the greatest single diameter.

# 17.2.2.2 Systemic Reactions – Measurement and Evaluation

Systemic reactions include fever, nausea/vomiting, headache, fatigue, myalgia (muscle pain), arthralgia (joint pain) and rash will be reported in a standardized manner over a period of 10 consecutive days after vaccination.

Systemic reactions will be rated based on the FDA Guidance on Toxicity Grading Scales as described in Table 17.2-2. Any grade 4 systemic reaction should be reported as an SAE (see Section 17.1.2).

Induration / swelling should be evaluated and graded using the functional scale as well as the actual measurement.

e Any Grade 4 injection site reaction will be reported as SAE, Grade 3 severity should be documented.

Table 17.2-2 Grading of Systemic Reactions - Vaccine Specific Criteria Potentially Life Vaccine-specific Mild Moderate Severe Threatening (Grade 4) d Criteria (Grade 1) (Grade 2) (Grade 3) 38.0 - 38.4 °C 38.5 - 38.9 °C 39.0 - 40.0 °C > 40.0 °C Fever a 100.4-101.1 °F 101.2-102.0 °F 102.1-104 °F >104 °F No interference Prevents daily Some interference ER visit or with activity or 1 activity, requires Nausea/vomiting with activity or > 2 hospitalization for 2 episodes/24 outpatient IV episodes/24 hours hypotensive shock hours hydration Repeated use of non-narcotic pain Significant; any use No interference reliever > 24 hours of narcotic pain ER visit or Headache with activity or some reliever or prevents hospitalization daily activity interference with activity No interference Some interference Significant; prevents ER visit or **Fatigue** with activity with activity daily activity hospitalization No interference Some interference Significant; prevents ER visit or Myalgia with activity with activity daily activity hospitalization No interference Some interference Significant; prevents ER visit or Arthralgia b with activity with activity daily activity hospitalization Macules/papules Macules/papules covering 10-30% Macules/papules covering <10% BSA with or without covering >30% BSA body surface area with or without symptom (e.g., Rash c (BSA) with or pruritus, burning, associated without symptoms symptoms; limiting tightness); limiting (e.g., pruritus, instrumental self care activity of burning, tightness) activity of daily daily living living

#### 17.2.2.3 Body Temperature Measurement

From vaccination (Day 1) until Day 11 after vaccination (i.e., the first 10 post-vaccination days including the day of vaccination), the subject should measure his/her body temperature orally once every evening , assessments by the subject should occur at the same time each day, starting approximately 8 hours after vaccination. To optimize the comparability of the documented body temperatures, all subjects will be provided with a digital oral thermometer and be instructed in its use. The subjects may keep the thermometer after study termination.

<sup>&</sup>lt;sup>a</sup> Oral temperature; no recent hot or cold beverages or smoking.

<sup>&</sup>lt;sup>b</sup> Symptom not described in FDA Toxicity Grading Scale.

<sup>&</sup>lt;sup>c</sup> Grading based on Common Terminology Criteria for Adverse Events (CTCAE), NIH, v4.03, 2010.

d Any Grade 4 systemic reaction will be reported as SAE, Grade 3 severity should be documented.

If fever (oral body temperature  $\geq 38.0$  °C/100.4 °F) occurs, body temperature should be measured at least every 4 to 8 hours until it returns to normal (< 38.0 °C/100.4 °F). All body temperature measurements including the date and time should be recorded in the Subject eDiary (see Section 17.3). In case of fever, the subject should record all fever measurements in the diary including the first value that shows a return to normal body temperature.

Body temperature measurements from vaccination (Day 1) until Day 11 after vaccination (i.e., the first 10 post-vaccination days including the day of vaccination) will be transcribed automatically or by the Investigator into the eCRF. If more than one body temperature value is recorded in the diary for a given day, the highest daily temperature reading will be recorded in the eCRF.

Body temperature measurements will be analyzed according to the FDA Guidance on Toxicity Grading Scales for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (Food and Drug Administration) for data analysis as described in **Table 15.2-2** above.

Outside of the first 10 post-vaccination days, daily body temperature measurement is **not required**. However, subjects experiencing an AE with symptoms of fever are recommended to measure their body temperature in order to document fever as an AE in the eMemory Aid. If fever (i.e., oral body temperature ≥38.0°C/100.4 °F) occurs, it is recommended that the subject measures his/her body temperature every 4 to 8 hours until fever resolves (i.e., oral body temperature <38.0°C/100.4 °F) in order to document onset and resolution, as defined by the date of first oral body temperature measurement of ≥38.0°C/100.4 °F (date of onset) and the date of first oral body temperature measurement of <38.0°C/100.4 °F (date of resolution).

### 17.3 Study eQuestionnaires

Subjects will be provided with two types of electronic questionnaires throughout the course of this study:

- > Subject eDiary will be distributed to all subjects for the collection of safety information from the day of vaccination until the first 10 post-vaccination days (i.e. including the day of vaccination)
- ➤ eMemory Aid will be distributed to all subjects for the collection of safety information outside the first 10 post-vaccination days until the next Visit .

The following information will be collected in the Subject eDiary (10 days post-vaccination):

- Measurement of oral body temperature (For further information see Section 17.2.2.3);

- Solicited injection site reactions <sup>xii</sup> (injection site pain, tendemess, redness, induration and swelling), for further information see Section 17.2.2.1;
- Solicited systemic reactions xii (fever, fatigue, headache, nausea/vomiting, muscle pain, joint pain, rash);
- Other AEs:
- Any new concomitant medication or changes in medication taken after vaccination;
- Information on travel to geographical regions where CHIKV is endemic.

The following information will be collected in the eMemory Aid (outside 10 day post-vaccination period):

- AEs:
- Any new concomitant medication or changes in medication taken after vaccination;
- Ongoing solicited reactions;
- Information on travel to geographical regions where CHIKV is endemic.

Assessments by the subject should occur at the same time each day, starting approximately 8 hours after vaccination. The subject will be properly instructed on the reporting requirements and how to complete and use the subject diaries, thermometer and measuring device (for assessment of measurable injection site reactions).

Questionnaires are always to be assessed at the next visit by the Investigator together with the subject, prior to these data being entered into the electronic case report form (eCRF). The Investigator will review and discuss the questionnaires with the subject, ask about AEs occurring since the last visit and ensures completeness and reliability of self-reporting. The entries in the respective questionnaires shall be evaluated and graded for severity and relatedness to the vaccination by the Investigator.

The eQuestionnaires will serve as source documentation. Entries in the eQuestionnaires will be transcribed into the appropriate eCRFs. Any entry on the eCRF that does not correspond with an entry in the eDiary will be explained by the Investigator on the relevant questionnaire page.

# 17.4 Medical, Medication, and Non-Drug Therapy History

#### 17.4.1 Medical history

At screening, the subject's medical history will be described for the following body systems including severity (mild, moderate, or severe as defined in Section 17.2.1.1) or surgery and

xii Solicited injection site and systemic reactions in the Subject eDiary will be assessed by the subject for absence, presence and duration.

start and end dates, if known: eyes, ears, nose, and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological; endocrine; metabolic; hematopoietic/lymphatic; dermatological; and genitourinary.

In addition, the medical history covering the last 3 years prior to screening will include the following:

- Information on prior vaccination against relevant traveler diseases (i.e. yellow fever, Japanese encephalitis)
- Previous chikungunya virus infection;
- Other vector-borne diseases in the past;
- Previous trauma to joints;
- Information on planned hospitalizations (including elective surgery) during the study for medical conditions existing prior to or at study entry. Such planned hospitalizations will not need to be reported as SAEs.

# 17.4.2 Concomitant Medications and Non-Drug Therapies

All medications (including vaccinations) received from 2 weeks prior to study enrollment until completion/termination should be collected from all subjects, and recorded on the appropriate eCRF. In addition to product name (generic name), the dose, indication, route of administration and frequency as well as the start and end date of treatment will be documented.

In addition, medications to treat SAEs will be reported to the Sponsor on SAE Report Forms as described in Section 3. In context of this study, information on non-drug therapies will only be collected in relation to SAEs.

The following medications are **not permitted** if administered within the specified study periods (unless such treatment has to be administered in an emergency situation):

- Any blood products or immunoglobulins during the course of the study;
- Immunosuppressive therapies (e.g. systemic or high dose inhaled [>800 μg/day of beclomethasone dipropionate or equivalent] corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs) during the course of the study;
- Prophylactic administration of antipyretics within 4 hours prior to and during the first 72 hours after vaccination;
- > Subjects are requested to refrain from donation of blood, blood fractions and plasma within 30 days prior to vaccination and for the entire study duration

For documentary purposes, any of the treatments listed above (including emergency treatment) given within these time periods requires special documentation and is to be documented as a protocol deviation.

The following medications and procedures will delay vaccination:

- antipyretics received within 4 hours prior to vaccination.
- any live or inactivated vaccine received within 28 days or 14 days prior to vaccination, respectively.

Usage of any other medications or non-drug therapies is not restricted.

Additionally, medications that are not permitted prior to study enrollment, resulting in exclusion from the study, are reflected in the exclusion criteria in Section 13.2.

### 17.5 Vital Signs

Vital signs will include body temperature (°C / °F) measured orally, pulse rate (beats/min), and systolic and diastolic blood pressure (mmHg) while seated and at rest.

Vital signs will be measured at screening (Visit 0) and at the vaccination visit (Visit 1) and are to be recorded before the vaccination is given. In addition, after an observation period of 30 minutes at the study site following vaccination pulse rate as well as blood pressure while seated and at rest will again be assessed.

Vital sign values are to be recorded on the appropriate eCRF. For each vital sign value, the Investigator will determine whether the value is considered an AE (see definition in Section 17.1.1). If assessed as an AE, the medical diagnosis (preferably), symptom, or sign, will be recorded on the AE eCRF. Additional tests and other evaluations required to establish the significance or etiology of an abnormal result, or to monitor the course of an AE should be obtained when clinically indicated. Any abnormal value that persists should be followed at the discretion of the Investigator.

#### 17.6 Physical Examinations

At screening (Visit 0), a physical examination will be performed on the following body systems being described as **normal** or **abnormal**: general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, skin, and neurological.

A symptom-driven physical examination will be performed at all study Visits except the Screening Visit (Visit 0), i.e. only in case a symptom is reported by the subject, a system-based assessment will be performed for a detailed check of the affected body system(s). A symptom-driven examination should also be performed in case the subject has complaints within the observation time after vaccination (as described in 24.2, Visit 0 Screening).

A Hand Stiffness examination will be performed at all study Visits irrespective of any clinical signs or symptoms. The subject will be asked to bend simultaneously the four fingers of both hands, i.e. index, middle, ring, and little finger and the range of motion will be measured with a measuring device. Specifically, the distance between the fingers and

the ball of the thumb should be measured in cm or inch. The distance of the least flexible finger of each hand should be measured and recorded in the eCRF. Importantly, the same finger of each hand should be measured for subsequent visits. Special attention should be paid to measuring consistently to the same part of the ball of the thumb.

Abnormal conditions detected at screening or prior to vaccination at Visit 1 will be recorded as medical history. At all other study visits, if a new abnormal or worsened abnormal preexisting condition is detected, the condition will be recorded as an AE. A quidance document on the hand stiffness test is included in the Supplement Section (see Section 24.4).

# 17.7 Clinical Laboratory Parameters

Blood and urine samples will be obtained for assessment of clinical laboratory parameters as outlined in the Schedule of Study Procedures (see Section 24.2) or in the Screening and Study Visits Section (see Section 15.4). Parameters will be analyzed by central laboratories according to the applicable laboratory SOP.

# 17.7.1 Safety Sample

A (baseline) safety laboratory blood [13.0 mL] and urine sample will be obtained at Visit 0 (Screening Visit) and all subsequent visits from all subjects for standard clinical chemistry. hematology, coagulation panel and urinalysis as well as for HIV / HBsAg / HCV [5.0 mL] testing (at the Screening Visit only).

sodium,

potassium.

Creatinine,

| Clinical chemistry (approx. 3.5 mL) | Creatinine, sodium, potassium, calcium, aspartate transaminase (AST), alanine aminotransferase (ALT), alkaline phosphatase, bilirubin and C-reactive protein (CRP). |
|---|---|
| Hematology panel (approx. 5.0 mL) | Hemoglobin, hematocrit, erythrocyte count, WBC count, differential WBC count (basophils, eosinophils, lymphocytes, monocytes, neutrophils), platelets, ESR. |
| Coagulation panel (approx. 4.5 mL) | Small blood coagulation (prothrombin time, aPTT and fibrinogen). |
| HBsAg/ HCV / HIV test<br>(approx. 5.0 mL) | A positive HIV test obtained by ELISA will have to be confirmed by a second method [e.g. Western blotting or PCR], at Visit 0 only. |
| <u>Urinalysis</u> | Standard urine dipstick for determining pH-value, specific gravity, leucocytes, nitrite, protein, glucose, ketones, |

urobilinogen, bilirubin, erythrocytes.

## 17.7.2 CHIKV Screening

A CHIKV baseline Screening Sample (5.0 mL) will be obtained from ALL subjects at Visit 0 (Screening Visit) for CHIKV-specific ELISA testing for subjects by baseline serostatus.

### 17.7.3 COVID-19 Sample

A COVID-19 Sample [5.0 mL] will be obtained from all subjects at Visit 1 (Day 1), Visit 3 (Day 29), Visit 5 (Day 180) and at the ET for retrospective serological Sars-CoV-2 specific antibody testing.

### 17.7.4 Baseline Sample

A Baseline Sample [10.0 mL] will be drawn from all subjects at Visit 1 (Day 1) for retrospective investigation of potential pre-existing antibodies including but not limited to other alphaviruses (i.e. Mayaro), dengue or Zika. Such assessments may occur at laboratories other than the central laboratory used for analysis of safety samples.

### 17.7.5 Assessment of Laboratory Values

Laboratory values will be evaluated according to the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (Food and Drug Administration). For the individual toxicity criteria refer to Section 24.3.

Laboratory assessments for which no severity grading is described in Section 24.3 are graded as described in Section 17.2.1.1 upon investigator's judgment.

The Investigator's assessment of each abnormal laboratory value, including its clinical significance, is to be recorded in the eCRF:

- Abnormal laboratory assessments that are considered clinically relevant, in the opinion of the Investigator, need to be documented as unsolicited AEs and assessed further for severity according to the toxicity grading scale provided in Section 24.3, causality and other assessments done for unsolicited AE (see Section 17.2.1).
- Abnormal laboratory assessments that are considered a symptom of an underlying AE or part of a syndrome that is reported as AE (e.g. presence of blood cells in urine in a person diagnosed with urinary tract infection) do NOT additionally need to be documented as unsolicited AE, but a respective comment should be added to the underlying AE.

Additional tests and other evaluations required to establish the significance or etiology of an abnormal laboratory result, or to monitor the course of an AE should be obtained when clinically indicated. Any abnormal value that persists should be followed at the discretion of the Investigator.

#### 17.8 Viremia

Subjects will return to the study site to collect plasma samples from all subjects on the vaccination Day 1 and on Days 8 and 29 (Visit 1-3), and if applicable at the ET Visit. Viremia plasma sample will be obtained from all subjects for a clinically indicated retrospective investigation of viremia by quantitative RT-PCR (RT-qPCR). The retrospective analysis will be conducted if deemed necessary by the Data Safety Monitoring Board upon clinical indication.

Viremia will be analysed in plasma samples. Blood [8.0 mL] will be collected by venous puncture. Samples will be shipped on dry ice at -70°C, viral RNA will be isolated and viral CHIKV RNA will be amplified specifically by RT-gPCR.

# 17.9 Adverse Events of Special Interest (AESI)

In addition to nonspecific transient muscle pain and joint pain that may occur after vaccination with any vaccine, subjects will be carefully monitored for signs and symptoms suggesting an acute stage CHIKV-associated event.

If a subject develops symptoms suggestive of CHIKV infection, he/she will be asked to contact the site immediately for clinical evaluation at an unscheduled visit.

Therefore, the following cluster of symptoms with or without remissions or exacerbations will receive particular consideration:

1. Fever (≥ 38.0 °C / 100.4 °F measured orally);

AND

2. Acute (poly)arthralgia/arthritis most frequently in the extremities (wrists, ankles and phalanges, often symmetric), back pain and/or neurological symptoms (e.g. confusion, optic neuritis, retinitis/uveitis meningoencephalitis or polyneuropathy) and/or cardiac symptoms (e.g. myocarditis);

OR

One or more of the following signs and symptoms: macular to maculopapular rash (sometimes with cutaneous pruritus (foot arch) and edema of the face and extremities), polyadenopathies;

AND

3. Onset of symptoms 2 to 21 days after vaccination;

AND

4. Duration of event ≥ 3 days.

Any suspected clinical case of CHIKV-associated event shall be referred to a clinical expert, be evaluated according to standard diagnostic procedures and treated according to current medical standard until resolved or stabilized. For more detailed information please refer to: French guidelines for the management of chikungunya - acute and persistent presentations (Simon, Javelle et al. 2015).

Additionally, subjects presenting with acute arthralgia within 2 to 21 days post-vaccination will be followed-up until resolution and monitored for recurrences until the end of the study.

A blood sample for laboratory investigation will be taken upon presentation of the subject. Testing may include but is not limited to rheumatoid factor (RF), anticitrullinated protein antibody (ACPA), Ferritin and CRP. Retrospective investigation of a pre-vaccination sample may be considered for a thorough causality assessment.

Suspected CHIKV-associated events do not constitute a reason for withdrawal from the study.

#### 17.10 Adverse Event Reporting Procedures

#### 17.10.1 Serious Adverse Event

Any SAE should be reported to the Safety Desk by fax or email within 24 hours after the Investigator has become aware of the event. Under certain circumstances the initial notification could be done by phone, but nevertheless a written SAE Report Form has to be submitted to the Safety Desk within 24 hours (see Section 3).

Correct SAE reporting will have to cite a diagnosis or a symptom. Any diagnosis and any symptom is regarded as separate SAE. However, if the Investigator considers several symptoms to be in the context of one underlying diagnosis, he/she may specify the diagnosis as the reportable SAE and describe the attendant symptoms in one single appropriate SAE report.

Medical or diagnostic procedures due to an underlying disease or symptom are not considered an AE but a consequent measure following an AE. A correct SAE report will therefore have to specify the disease or symptom as the reportable AE and the medical or diagnostic procedure as action taken.

In addition, expedited and periodic reporting to Competent Authorities and IRBs will be performed in accordance with local requirements. Further reporting details can be found in the study-specific SAE procedure which is in accordance with respective US/EU requirements, International Conference on harmonization (ICH) GCP, national laws and site-specific requirements. SAEs that are considered as probably or possibly related and additionally are unexpected need to be reported according to the requirements for suspected unexpected serious adverse reactions (SUSARs).

SAE reports will be reviewed by a study site's physician, the Safety Desk, the Study Medical Monitor, the Sponsor and the independent DSMB.

Beyond study end, if the investigator becomes aware of SAEs that are fatal, life-threatening or suspected to be related to study treatment will continue to be reported until 6 months after the last study visit of the respective subject (i.e. Visit 5).

# 17.10.2 Adverse Events of Special Interest (AESI)

Any AESI should be reported to the Safety Desk by fax or email within 48 hours after the Investigator has become aware of the event. Under certain circumstances the initial notification could be done by phone, but nevertheless a written AESI Report Form has to be submitted to the Safety Desk within 48 hours (see Section 4).

Subjects will be carefully monitored for development of AESIs. A cluster of symptoms (see 17.9) associated with CHIKV infection, are defined as AESI. In case an AESI is identified, the Investigator will complete the AESI Report Form with all available information including medical records. This information will be provided to the DSMB. The DSMB will perform a thorough review of each case and advise whether additional clinical work-up is required.

The DSMB will conduct a final adjudication of all AESIs and will assess whether cases were new in onset and whether there is any relationship to administration of the study vaccine. Narratives with detailed case descriptions will be provided for all AESIs.

#### 17.10.3 Pregnancy

The risk of maternal to fetal transmission of chikungunya virus during pregnancy cannot be excluded. Thus, women must not become pregnant during the first three months post-vaccination.

Reporting requirements start with administration of the vaccination until study completion (or ET Visit). All pregnancies that occur during the clinical study period will be followed-up for three months after delivery or termination of the pregnancy. Any effect on either mother or fetus should be determined. A pregnancy which led to a congenital anomaly/birth defect must be followed-up by the Investigator longer or until resolution or stabilization. Duration of prolonged follow-up will be decided on an individual basis and in accordance with the Sponsor. The Investigator will prepare a narrative on the course of the pregnancy and the outcome.

The Investigator should report pregnancies within 24 hours of being notified using the Pregnancy Report Form. Reporting procedures are similar to SAE reporting procedures (contacts and processing), although a pregnancy is not considered an SAE (see Section 5).

If a seriousness criterion applies in addition to the pregnancy (e.g. hospitalization, congenital anomaly/birth defect) the pregnancy qualifies as an SAE. In such case a Pregnancy Report Form and an SAE Report Form have to be filled out.

### 17.11 Safety Monitoring

# 17.11.1 Data Safety Monitoring Board

An independent Data Safety Monitoring Board (DSMB) will be utilized for this study. The DSMB will consist of four voting members who will be selected based upon their expertise with and understanding of infectious diseases, vaccines, clinical research and/or skills and knowledge in clinical medicine. The DSMB will meet to review accumulating safety data on a regular basis until all subjects have received the vaccination at Day 1 and until all subjects have completed Visit 2 or 3. In addition, the DSMB will periodically review accruing safety information throughout the study, as applicable. A meeting of the DSMB may be called at the discretion of the Sponsor, e.g. to address any safety concerns arising during the conduct of the study.

The DSMB will ad hoc review cases of SAEs, AESIs and severe (Grade 3) solicited AEs. The DSMB will periodically review listings and summary tabulations of SAEs, Deaths, Solicited AEs, Unsolicited AEs.

A DSMB charter including a detailed description will be prepared.

#### Responsibilities of the DSMB

- Provides independent monitoring of safety issues, which means it reviews and evaluates all SAE reports and study discontinuations for: (i) increases in frequency of SAEs and study discontinuations within the study; and (ii) SAEs in the study sample compared with the population based on what is known from the literature;
- Reviews data produced from the study upon the Sponsor's request to determine whether the conditions on which study design is based have remained the same or have changed. If changed, the DSMB will suggest whether or not the changes mandate changes to the protocol and suggest a protocol amendment;
- Upon the Sponsor's request, meets for discussion and gives recommendations to the Sponsor as to whether the study should progress unchanged, or the study requires changes, or the study should be terminated prematurely;
- > Can propose an unplanned safety analysis of clinical trial data;
- Can suggest unscheduled visits for specific evaluations for individual cases reviewed.

# 17.11.2 Sponsor

Until the last subject reached Day 29, listings of available blinded safety data will be closely reviewed by the Sponsor to identify any potential safety concerns.

# 17.11.3 Investigator

To ensure information exchange on safety across sites, Investigators will be provided with safety information pertaining to all severe (Grade 3) AEs and SAEs reported in the eCRF.
### 18. STATISTICS

### 18.1 Sample Size Justification

The sample size is selected to allow for a demonstration of Lot-to-Lot consistency based on the primary endpoint, CHIKV-specific neutralizing antibody titers as determined by microneutralization (µPRNT) assay on Day 29 post-vaccination. The primary analysis will demonstrate equivalence between the three treatment groups based on a comparison of GMTs.

402 randomized subjects (i.e. 134 per batch) will ensure that the three pair-wise comparisons have an overall power of approximately 90% based on a two-sided significance level of 5%, an assumed SD of 0.32 (on a log10 scale), and acceptance margins of the GMT ratios, while correcting for an assumed drop-out rate of 10%, 5% of subjects with major protocol deviations and 2% expected to be baseline positive for CHIKV.

### 18.2 Datasets and Analysis Cohorts

The full analysis set contains all subjects who were randomized and received at least one vaccination. Subjects will be analyzed as randomized.

The safety analysis set contains all subjects who entered into the study and received at least one vaccination. Subjects will be analyzed as treated.

The per protocol (PP) analysis set contains all subjects who were baseline negative for CHIKV antibodies and have received the vaccination and have evaluable immunogenicity data at baseline and the time point for the primary endpoint without a major protocol violation. Examples that may lead to exclusion from the PP population are provided here, further criteria may be defined in the Statistical Analysis Plan (SAP):

Subject has a known or suspected defect of the immune system that can be expected to influence the immune response to the vaccine, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to Visit 1. Immuno-suppressive therapy is defined as administration of chronic (longer than 14 days) prednisone or equivalent ≥ 0.05 mg/kg/day within 4 weeks prior to study entry, radiation therapy or immunosuppressive cytotoxic drugs/ monoclonal antibodies in the previous 3 years; topical and inhaled steroids are allowed;

- Subject is positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
- > Subject has received the wrong (not according to randomization) or no IMP.

These criteria for protocol violations are identified at the time of planning the study. However, during the course of the trial unforeseen events may occur or new scientific knowledge may become available, therefore final decisions on whether a protocol violation could impact on the immune response and thus lead to exclusion from the PP population will be made by the sponsor on a case by case basis in a blinded manner (prior to study unblinding). Sample testing issues may also lead to exclusion from the PP analysis for particular time points.

### 18.3 Handling of Missing, Unused, and Spurious Data

All statistical analysis will generally be based on observed values, missing values will not be imputed. In case of >5% of missing values for an immunogenicity comparison involving a statistical test, multiple imputation methods will be applied in order to evaluate the possible impact of missing values on these results.

### 18.4 Methods of Analysis

A statistical analysis plan will be prepared before database closure/snapshot.

### 18.4.1 Primary Endpoint

The primary immunogenicity analysis will be a comparison of the GMTs in the per-protocol (PP) analysis set between the VLA1553 Lots 1, 2 and 3 at Day 29 (i.e. 28 days post-vaccination) by ANOVA (factor Lot, covariate study site). The ANOVA model will be applied to the log10-transformed µPRNT values of the three Lots and the 95% CIs for the pair-wise ratios of the GMTs will be obtained by taking the anti-log of the resulting 95% CIs for the least square means differences. If these three pairwise 95% CIs for GMT ratios are all between equivalence between the three commercial batches will be postulated.

The analysis will be performed on the PP population who were baseline negative for CHIKV antibodies and will be repeated on the full analysis set.

### 18.4.2 Secondary Endpoints

### 18.4.2.1 Secondary Safety Endpoints

Safety tabulations will generally be provided separately for solicited AEs and unsolicited AEs, and for both types of AEs combined. 95% confidence intervals according to Altman will generally be provided for all AE rates and differences between the three Lots will be

assessed for significance using Fisher's exact test. Further details in addition to the outline below will be provided in the SAP.

The number and percentage of subjects with any AE, any solicited AE, unsolicited AE, any related unsolicited AE, any related severe AE, any SAEs, any related SAEs, any AESI, any related AESI, any medically attended AE, any AE leading to withdrawal from study, and any AE occurring at a frequency of at least 10% and at least 1% in at least one treatment group, up to Day 29, and up to Month 6, will be presented for each Lot overall and by system organ class/preferred term. Differences between the Lots will be assessed for significance using Fisher's exact test, a significant overall test will be amended by pair-wise tests.

Changes in laboratory values from study entry will be analyzed descriptively and will be part of the unsolicited AE evaluation only in case of clinically relevant deviations. The rates of subjects with laboratory assessments outside the normal range, and with abnormal laboratory parameters falling into the grade 0 vs. 1 through 3 will be calculated by visit and overall. The rate of subjects with urinalysis results according to the test manufacturer's results categories will be calculated.

All subjects entered into the study, who receive the single vaccination, will be included in the safety analysis.

### 18.4.2.2 Secondary Immunogenicity Endpoints

Secondary immunogenicity analysis will include the comparison of the GMTs between the three Lots at Day 8, Day 85 and Month 6 post-vaccination by ANOVA (factor Lot and covariate study site), two-sided 95% confidence intervals will be calculated for the GMT; GMFIs will be analyzed as outlined for GMTs. In addition, the seroprotection and seroconversion rates for various study days, and when applying other threshold titers for defining seroconversion or seroprotection thresholds will be compared between the treatment groups by Fisher's exact test and 95% confidence intervals will be calculated.

Analysis will be performed on the PP analysis set. It will be specified in the SAP which secondary immunogenicity analysis will be repeated for the full analysis set.

### 18.5 Planned Data Analysis of the Study

The following data analyses will be performed:

- Part A includes immunogenicity and safety data after all subjects have completed Visit 3 (Day 29);
- Part B includes immunogenicity and safety data after all subjects have completed Visit 5 (Month 6).

Individual study parts will be analyzed sequentially.

The Part A analysis will be performed once the last subject has completed the study Visit 3 (Day 29). Part B analysis will be performed once the last subject has completed the study Visit 5, i.e. Month 6, respectively. Part A will be unblinded but blind will be maintained for study sites.

### 19. ETHICS AND REGULATORY ASPECTS

### 19.1 Compliance Statement

This study will be conducted in accordance with this protocol, current ICH/GCP guidelines, Declaration of Helsinki, and with the applicable national and local regulatory requirements.

### 19.2 Institutional Review Board (IRB) and Regulatory Authorities

Before enrollment of healthy volunteers into this study, the protocol, informed consent form, any promotional material/advertisements, and any other requested information will be reviewed and approved/given favorable opinion by the IRB and applicable regulatory authorities in accordance with local requirements. The study will commence only upon the Sponsor's receipt of approval/favorable opinion from the IRB.

If the protocol and/or any other information given to the subject is/are amended, the revised document(s) will be reviewed and approved/given favorable opinion by the IRB and applicable regulatory authorities in accordance with local requirements, where applicable. The protocol amendment will only be implemented upon the Sponsor's receipt of approval. Amendments that are intended to eliminate an apparent immediate hazard to subjects may be implemented prior to receiving IRB and authority approval. However, in this case, approval must be obtained as soon as possible after implementation.

### 19.3 Subject Information and Informed Consent

It is the Investigator's responsibility to obtain freely given written informed consent from the subject before the subject is exposed to any study-related procedures, including screening tests for eligibility.

The informed consent form will include a comprehensive explanation of the proposed treatment without any exculpatory statements, in accordance with the elements required by ICH GCP and applicable regulatory requirements. Volunteers will be allowed sufficient time to consider participation in the study after having the nature and risks of the study explained to them. By signing the informed consent form, volunteers agree that all evaluations required by the study will be completed, unless they withdraw voluntarily or are terminated from the study for any reason.

The Investigator will explain that the subjects are completely free to refuse to enter the study or to withdraw from it at any time, without any prejudice and need for justification.

The subjects will be informed that representatives of the Sponsor and health authority inspector may review their source records, and that these persons are bound by confidentiality obligations.

The subject will be given a copy or a second original of the ICF. An original of the signed and dated ICF must be retained in the site's records, and is subject to inspection by representatives of the Sponsor or representatives from regulatory agencies.

The Sponsor will provide to the Investigator in written form any new information that significantly bears on the subjects' risks associated with study vaccine exposure. The informed consent form will be updated, if necessary. This new information and/or revised informed consent form, that has been approved by the applicable IRB and regulatory authorities, where applicable, will be provided by the Investigator to the subjects who consented to participate in the study.

### 20. QUALITY CONTROL AND QUALITY ASSURANCE

### 20.1 Source Data and Records

Source data are defined as all information related to clinical findings, observations or other activities in the study, captured in original records or certified copies of original records. The Investigator will permit study-related monitoring, audits, IRB review and regulatory inspections, by providing direct access to source data/records. Source records should be preserved for the maximum period of time required by local regulations.

Source data entries must be made in accordance with local requirements. Signed and dated copies of the laboratory result reports have to be kept within the subject's source data file.

eCRFs will not be used as source data for any other variable.

### 20.2 Investigator's Responsibility

The Investigator will comply with the protocol (which has been approved/given favorable opinion by the IRB), ICH GCP, and applicable regulatory requirements. The Investigator is ultimately responsible for the conduct of all aspects of the study at the study site and verifies by signature the integrity of all data transmitted to the Sponsor. The term "Investigator" as used in this protocol, and in study documents refers to the Investigator or authorized study personnel whom the Investigator has designated to perform certain duties. Sub-investigators or other authorized study personnel are eligible to sign for the Investigator, except where the Investigator's signature is specifically required.

### 20.3 Training

The study monitor will ensure that the Investigator and study site personnel understand all requirements of the protocol, the investigational status of the vaccine, and his/her

regulatory responsibilities as an Investigator. Training may be provided at an Investigator's meeting, at the study site, and/or by instruction manuals. In addition, the study monitor will be available for consultation with the Investigator and will serve as the liaison between the study site and the Sponsor.

### 20.4 Monitoring

A designated monitor will check electronic system data and source data at regular intervals throughout the study to verify completeness, accuracy and consistency of the data, protocol adherence, and adherence to GCP guidelines. The monitor will work and perform Source Data Verification according to the Clinical Management Plan. The Investigator will cooperate with the monitor to ensure that any discrepancies identified are resolved.

### 20.5 Audit and Inspection

Upon request, the Investigator will make all study-related source data and records available to a qualified quality assurance auditor mandated by the Sponsor or to regulatory inspectors. The main purposes of an audit or inspection are to confirm that the rights and welfare of the subjects have been adequately protected, and that all data relevant for the assessment of safety and efficiency of the investigational product have appropriately been reported to the Sponsor.

### 20.6 Non-compliance with the Protocol / Protocol Deviations from the Protocol

Any deviations from the protocol will be tracked, actions defined, as feasible, and reviewed in Data Review Meetings for the study part analysis and the final analysis for assessment of their influence on the quality of the study analysis.

### 20.7 Confidentiality of Subject's Data

The Investigator will exercise all reasonable precautions within the constraints of the applicable regulatory requirements to maintain the confidentiality of subjects' identities. On exported electronic source data or any other documents submitted to the Sponsor, subjects will only be identified by subject number. Documents not for submission to the Sponsor, e.g. subject identification log and original ICF, will be maintained by the Investigator in strict confidence.

### 21. DATA HANDLING AND RECORD KEEPING

### 21.1 Information of Investigators

An IB containing all important data relating to the safe use of the IMP will be supplied to the Investigator prior to study start.

The Investigator will be kept informed on new relevant safety data as the study proceeds.

### 21.2 Electronic Case Report Forms (eCRFs)

### 21.2.1 Data Recorded Directly on Case Report Forms

An electronic Case Report Form (eCRF) will be used for this study. Data will be recorded directly onto source documents before documentation in the eCRF.

### 21.2.2 eCRF entries

eCRF entries and corrections will only be performed by study site staff authorized by the Investigator. Each user is informed of the clinical study's web-site internet address and is allocated to a user account with personal password to access the confidential website. The personal password must be kept confidential and must only be used by the person to whom it was assigned. For additional authorized users at the site, a new user account has to be requested to ensure that each entry/change can be allocated to the person who performed the entry/change.

All visit data need to be recorded in the eCRF database as soon as possible after each study visit, no later than 1 business day after data has been collected.

### 21.2.3 Changes to eCRF data

Corrections may be requested as follows:

- ➤ Investigators' responses are checked as they are entered and are rejected if they do not fulfill quality criteria. A message will specify the type of error or syntax error and assist in its correction.
- > If required, the CRA can ask for information to be corrected during monitoring.
- Computerized data-check programs and manual checks will identify clinical data discrepancies for resolution. Corresponding queries will be created within the data capturing system and the site will be informed about new issues to be resolved online.

All discrepancies will be solved on-line directly by the Investigator or by authorized staff.

Corrections of eCRF data may be performed by authorized staff only. The person performing the changes in the eCRF is required to electronically confirm the changes made.

### 21.2.4 eCRF Entry Validation

The Investigator will thoroughly review the data on the eCRF, and will finally certify the contents of the eCRF by electronic signature after completion of each subject. If a correction is made to the eCRF data after the Investigator's final approval, the certification must be repeated after the changes have been performed.

### 21.2.5 Data collection

All visits and assessments are entered into an interactive form. eCRFs will be source document verified following guidelines established before study onset and detailed in the Monitoring Plan. Maintenance of the study database will be performed. Details to eCRF handling are provided in a study specific eCRF manual.

### 21.3 Coding of Adverse Events, Drugs and Diseases

After data entry, AEs and medical history will be coded according to the latest MedDRA version. The same MedDRA version will be applied to all study parts. Previous and concomitant medication and vaccines will be coded according to the latest version of the WHO Drug Reference List and Anatomical Therapeutic Chemical (ATC) Classification System.

### 21.4 Investigator File

### 21.4.1 Maintenance

The Investigator will maintain complete and accurate study documentation in a separate file (i.e. Investigator File) provided during the initiation visit. The Investigator is responsible for maintaining complete, up to date and accurate study records to enable the conduct of the study to be fully documented. The records should include the clinical protocol as well as any amendments, study approval letters, all original ICFs, drug dispensing and accountability logs and all relevant correspondence pertaining to the study.

### 21.4.2 Archiving and Destruction

All study-related documents should be kept by the Investigator for the maximum period of time required by local regulations. No study document should be destroyed without prior written agreement between the Investigator and the Sponsor. Should the Investigator elect to assign the study documents to another party, or move them to another location, the Sponsor must be notified.

### 21.4.3 Provision of Additional Information

On request, the Investigator will supply the Sponsor with additional data relating to the study or copies of relevant source records, duly anonymized. In case of particular issues or governmental queries, it is also necessary to have access to the complete study records, provided that the subject's confidentiality is protected in accordance with applicable regulations.

### 22. PUBLICATION POLICY

All results generated in this study will be considered to be strictly confidential. The Investigator may not submit the results for publication or presentation without prior written permission of the Sponsor. Authorship for any publication will be determined in mutual agreement. Within the scope of publication, co-authorship may be offered, at the sole discretion of the Sponsor, on a case by case basis taking scientific contribution into consideration. This is according to uniform requirements for manuscripts submitted to biomedical journals proposed by the International Committee of Medical Journal Editors.

### 23. LIABILITIES AND INSURANCE

In case of any damage or injury occurring to a subject in association with the participation in the study, insurance has been contracted.

The name, address and the insurance policy number will be given to both the Investigator prior to enrollment. Moreover a copy of the insurance conditions will be filed on site.

The Investigator is responsible for dispensing the investigational product according to this protocol, and for its secure storage and safe handling throughout the study.

page 82 / 90

24. SUPPLEMENTS

## 24.1 Study Flow Chart

Figure 24.1-1 Study Design for VLA1553-302



VLA1553

# 24.2 Schedule of Study Procedures and Assessments

Table 24.2-1 Schedule of Study Procedures and Assessments

| | | | PartA | | Part B | | ΞΞ |
|---|---|---|---|---|---|---|---|
| Procedures/Assessments | Visit 0<br>Screening<br>(Day -28 to<br>Day 0) | <b>Visit 1</b> <sup>m</sup><br>Day 1 | Visit 2<br>Day 8 | <b>Visit 3</b><br>Day 29<br>M1 | Visit 4<br>Day 85<br>M3 | Visit 5<br>Day 180<br>M6 | Visit |
| Informed consent a | × | | ļ | | | | |
| Inclusion/Exclusion criteria | × | X<br>(Review) | | | | | |
| Demographics <sup>b</sup> | × | | | | | | |
| Medical history <sup>e</sup><br>(including vaccination history) | × | X<br>(Update) | | | | | |
| Randomization | | × | | | | | |
| Prior/Concomitant medications | × | × | × | × | × | × | × |
| Physical examination and Hand Stiffness Test d | × | × | × | × | × | × | × |
| Vital signs e | × | × | | | | | |
| Baseline Sample f [10.0 ml] | | × | | | | | |
| CHIKV Screening ° [ 5.0, mL ] | × | | | | | | |
| COVID-19 Sample P [ 5.0 mL ] | | × | | × | | × | × |
| Serum/Urine Pregnancy test 9[3.0 mL] | × | × | | × | × | × | × |
| Immunogenicity h [40.0 mL] | | × | × | × | × | × | × |
| Safety Lab Sample [13.0 mL] | × | × | × | × | × | × | × |
| HIV / HBsAg / HCV testing [ 5.0 mL] | × | | | | | | |
| Viremia <sup>k</sup> [ 8.0 ml] | | × | × | X | | | × |
| VACCINATION | | × | | | | _ | |
| Subject eDiary | | | R | | | | R |
| eMemory Aid | | | l | R | R | Z. | ፚ |
| AE/AESI "/SAE Assessment | | × | × | × | × | × | × |

VLA1553

### ....instruct; R....review

- <sup>a</sup> Occurs at enrollment before Screening.
- <sup>b</sup> Demographics include year of birth, age, height, weight, BMI, gender, race and ethnicity
- Symptoms noted at Visit 1 (prior to first vaccination) are not considered AEs, but will be recorded as medical history. Prior vaccination against relevant traveler diseases should be documented in the Medical History, i.e. YF and JEV.
- general appearance, head and neck, eyes and ears, nose and throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, dat the screening visit, a physical examination will be performed on the following body systems being described as normal or abnormal: reported by the subject, a symptom-based assessment of the affected body system(s) will be performed. A hand stiffness and mobility skin, and neurological. At subsequent visits, a symptom-driven physical examination will be performed, i.e. only in case symptom is examination will be performed at all study visits irrespective of prior symptoms.
- e Vital signs will include systolic and diastolic blood pressure and pulse rate while seated and at rest, and body temperature measured orally before vaccination. In addition, after an observation period of 30 minutes following vaccination pulse rate as well as blood pressure while seated and at rest will again be assessed.
- f A baseline sample will be drawn for retrospective investigation of potential pre-existing antibodies including but not limited to e.g. a panel of alphaviruses (i.e. Mayaro) or dengue and Zika [blood (for all tests): 10.0 mL].
  - <sup>9</sup> A **serum** pregnancy test will be performed for all female subjects of childbearing potential at the screening visit only and a urine pregnancy test will be done prior to vaccination at Visit 1 and at indicated visits [blood: 3.0 mL].
    - analysis if deemed necessary by the Data Safety Monitoring Board upon clinical indication or on demand if requested later by regulatory Blood draw [40.0 mL] for CHIKV-specific neutralizing antibody titer evaluation, development of further assays or retrospective safety authorities
- aPPT, fibrinogen) and urinalysis (i.e. pH, specific gravity, leucocytes, nitrite, protein, glucose, ketones, urobilinogen, bilirubin, erythrocytes) alanine aminotransferase (ALT), alkaline phosphatase, bilirubin, CRP), hematology (i.e. Hemoglobin, hematocrit, erythrocyte count, white blood count, differential white blood cell count, platelets, erythrocyte sedimentation rate (ESR), coagulation panel (i.e. Prothrombin time, Safety laboratory sample for standard clinical chemistry (i.e. creatinine, sodium, potassium, calcium, aspartate aminotransferase (AST), IEDTA blood: 13.0 mLl
  - HIV / HBsAg / HCV testing will be only performed at the screening visit (Visit 0). A positive HIV test obtained by ELISA will have to be confirmed by a second method (e.g. Western blot or PCR) [blood (for all tests): 5.0 mL].
- conducted if deemed necessary by the Data Safety Monitoring Board upon clinical indication or on demand if requested later by regulatory Viremia plasma sample for clinically indicated retrospective investigation of viremia by RT-qPCR. The retrospective analysis will be authorities.
- Only if the ET visit occurs prior to Day 29, a viremia plasma sample should be obtained from the subject for clinically indicated retrospective investigation of viremia by RT-qPCR.
  - m All procedures/assessments (apart from Subject eQuestionnaire distribution and AE assessment) occur prior to vaccination (unless stated otherwise)
    - AESI assessment 2 to 21 days post-vaccination only.
- A CHIKV Screening Sample [5.0 mL] will be obtained at Visit 0 (Screening Visit) for CHIKV-specific ELISA testing for baseline serostatus. Test result remains valid for up to 60 days from sample collection.
- P A COVID-19 Sample [5.0 mL] will be obtained at Visit 1 (Day 1), Visit 3 Day 29), Visit 5 (Day 180) and at the ET for retrospective serological Sars-CoV-2 specific antibody testing

page 84 / 90

### 24.3 Toxicity Grading Scale for Abnormal Laboratory Assessments

| | Mild<br>(Grade 1) <sup>1</sup> | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life<br>threatening<br>(Grade 4) <sup>2,6</sup> |
|---|---|---|---|---|
| | Hematology Parameters | | | |
| Hemoglobin (Female) -<br>gm/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | <8.0 |
| Hemoglobin (Male) - gm/dL | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 | <8.5 |
| Hematocrit | Outside normal range <sup>3</sup> | | | |
| Erythrocyte count | Outside normal range <sup>3</sup> | | | |
| WBC Increase - cell/mm <sup>3</sup> | 10,800 – 15,000 | 15,001 – 20,000 | 20,001 – 25,000 | >25,000 |
| WBC Decrease - cell/mm <sup>3</sup> | 2,500 - 3,5004 | 1,500 - 2,499 | 1,000 – 1,499 | <1,000 |
| Neutrophils Decrease - cell/mm <sup>3</sup> | 1,500 – 2,000 | 1,000 – 1,499 | 500 – 999 | <500 |
| Lymphocytes Decrease - cell/mm <sup>3</sup> | 750 – 1,000 | 500 – 749 | 250 – 499 | <250 |
| Monocytes | | Outside no | rmal range <sup>3</sup> | |
| Eosinophils -<br>cell/mm³ | 650 – 1500 <sup>4</sup> | 1501 - 5000 | > 5000 | Hyper-<br>eosinophilic |
| Basophils | | Outside no | rmal range <sup>3</sup> | <u> </u> |
| Platelets Decreased - cell/mm <sup>3</sup> | 125,000 –<br>140,000⁴ | 100,000 –<br>124,000 | 25,000 – 99,000 | <25,000 |
| ESR | Outside normal range <sup>3</sup> | | | |
| | Clinical Chemistry Parameters | | | |
| Creatinine – mg/dL | 1.5 – 1.74 | 1.8 2.0 | 2.1 – 2.5 | >2.5 or requires dialysis |
| Sodium – Hyponatremia<br>mEq/L | 132 – 134 | 130 – 131 | 125 – 129 | <125 |
| Sodium – Hypernatremia<br>mEq/L | 144 – 1454 | 146 – 147 | 148 – 150 | >150 |
| Potassium – Hyperkalemia<br>mEq/L | 5.1 - 5.2 <sup>4</sup> | 5.3 – 5.4 | 5.5 – 5.6 | > 5.6 |
| Potassium – Hypokalemia<br>mEq/L | 3.5 – 3.64 | 3.3 – 3.4 | 3.1 – 3.2 | <3.1 |
| Calcium – Hypocalcemia<br>mg/dL | 8.0 - 8.44 | 7.5 – 7.9 | 7.0 – 7.4 | <7.0 |
| Calcium - Hypercalcemia mg/dL | 10.5 – 11.0 | 11.1 – 11.5 | 11.6 – 12.0 | >12.0 |
| AST increase by factor | 1.1 – 2.5 x ULN <sup>5</sup> | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | >10 x ULN |
| ALT – increase by factor | 1.1 – 2.5 x ULN | 2.6 - 5.0 x ULN | 5.1 – 10 x ULN | >10 x ULN |
| Alkaline phosphatase – | 1.1 – 2.0 x ULN | 2.1 – 3.0 x ULN | 3.1 10 x ULN | >10 x ULN |

| | Mild<br>(Grade 1) <sup>1</sup> | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially life<br>threatening<br>(Grade 4) <sup>2,6</sup> |
|---|---|---|---|---|
| increase by factor | | | | |
| Bilirubin – when<br>accompanied by any<br>increase in Liver Function<br>Test increase by factor | 1.1 – 1.25 x ULN | 1.26 – 1.5 x ULN | 1.51 – 1.75 x<br>ULN | >1.75 x ULN |
| Bilirubin – when Liver<br>Function Test is normal;<br>increase by factor | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| CRP | | Outside no | rmal range <sup>3</sup> | |
| | Coagu | ulation Factors | | |
| PT – increase by factor (prothrombin time) | 1.0 – 1.10 x<br>ULN <sup>5</sup> | 1.11 – 1.20 x<br>ULN | 1.21 – 1.25 x<br>ULN | > 1.25 ULN |
| PTT (aPTT) – increase by factor (activated partial thromboplastin time) | 1.0 – 1.2 x ULN | 1.21 – 1.4 x ULN | 1.41 – 1.5 x ULN | > 1.5 x ULN |
| Fibrinogen increase - mg/dL | 400 – 5004 | 501 – 600 | > 600 | |
| Fibrinogen decrease -<br>mg/dL | 150 – 2004 | 125 – 149 | 100 – 124 | < 100 or<br>associated with<br>gross bleeding or<br>disseminated<br>intravascular<br>coagulation (DIC) |

<sup>&</sup>lt;sup>1</sup> In case the laboratory's normal ranges and absolute Grade 1 limits overlap, Grade 1 limits will prevail, i.e. the value will be classified as Grade 1 abnormality even if it is within central laboratory normal ranges. Values between the central laboratory normal ranges and absolute Grade 1 limits will be reported as no abnormality (Grade 0).

<sup>&</sup>lt;sup>2</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as Potentially Life Threatening (Grade 4). For example, a low sodium value that falls within a grade 3 parameter (125-129 mE/L) should be recorded as a grade 4 hyponatremia unsolicited AE if the subject had a new seizure associated with the low sodium value.

<sup>&</sup>lt;sup>3</sup> As neither the FDA Scale nor the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (December 2004) provide any grading for Hematocrit, Erythrocyte count, Monocytes, Basophils, ESR and CRP, these will only be analyzed as "outside normal range", as determined by central laboratory standards and graded as described in Section 17.2.1.1 upon investigator's judgement

<sup>&</sup>lt;sup>4</sup> Central laboratory values should be adjusted to FDA toxicity grading scale. Specifically, if central laboratory reference range is more stringent than FDA toxicity grading scale the central laboratory values should be reported as no abnormality (Grade 0). Similarly, if laboratory values are within the central laboratory normal reference range, but fall into FDA toxicity grading scale, the values should be reported as indicated by the FDA toxicity grading scale.

<sup>&</sup>lt;sup>5</sup> "ULN" is the upper limit of the normal range.

<sup>&</sup>lt;sup>6</sup> Any grade 4 abnormal laboratory value should be reported as an SAE (see Section 17.1.2).

### 24.4 Guidance on Hand Stiffness Test

Please perform the Hand Stiffness Test at every study Visit on both hands irrespective of any clinical signs or symptoms. The subject will be asked to bend simultaneously the four fingers of both hands, i.e. index, middle, ring, and little finger and the range of motion will be measured with a measuring device. Special attention should be paid to measuring consistently to the same part of the ball of the thumb.

When measuring the distance in cm/inch between the fingers and the ball of the thumb, the distance between the ball of the thumb and the finger that is least flexible/mobile should be documented for the right and the left hand in the source document. At subsequent visits, the same least flexible finger of each hand should be measured and recorded in the source document.

Normal finger flexion:





Simulataneous finger flexion:





If the subject cannot bend fingers simultaneously, the distance in cm/inch between the ball of the thumb and the finger that is least flexible/mobile should be documented for the right and the left hand:



### 25. REFERENCES

- Ahola, T., T. Couderc, et al. (2015). "Therapeutics and vaccines against chikungunya virus." Vector Borne Zoonotic Dis **15**(4): 250-257.
- Broeckel, R., N. Haese, et al. (2015). "Nonhuman Primate Models of Chikungunya Virus Infection and Disease (CHIKV NHP Model)." <u>Pathogens</u> 4(3): 662-681.
- Chang, Lee Jah et al. 2014. "Safety and Tolerability of Chikungunya Virus-like Particle Vaccine in Healthy Adults: A Phase 1 Dose-Escalation Trial." The Lancet 384(9959): 2046–52. http://dx.doi.org/10.1016/S0140-6736(14)61185-5.
- Chen, Grace L. et al. 2020. "Effect of a Chikungunya Virus-Like Particle Vaccine on Safety and Tolerability Outcomes: A Randomized Clinical Trial." <u>JAMA Journal of the American Medical Association</u> 323(14): 1369–77.
- Couderc, T., N. Khandoudi, et al. (2009). "Prophylaxis and therapy for Chikungunya virus infection." J Infect Dis **200**(4): 516-523.
- Couderc, T. and M. Lecuit (2009). "Focus on Chikungunya pathophysiology in human and animal models." Microbes Infect 11(14-15): 1197-1205.
- Delisle, E., C. Rousseau, et al. (2015). "Chikungunya outbreak in Montpellier, France, September to October 2014." <u>Euro Surveill</u> **20**(17).
- Dubrulle, Mathieu et al. 2009. "Chikungunya Virus and Aedes Mosquitoes: Saliva Is Infectious as Soon as Two Days after Oral Infection." PLoS ONE 4(6).
- Edelman, R., C. O. Tacket, et al. (2000). "Phase II safety and immunogenicity study of live chikungunya virus vaccine TSI-GSD-218." Am J Trop Med Hyg **62**(6): 681-685.
- Food and Drug Administration, C. f. B. E. a. R. "Guidance for Industry: Toxicity Grading Scales for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials".
- Gorchakov, R., E. Wang, et al. (2012). "Attenuation of Chikungunya virus vaccine strain 181/clone 25 is determined by two amino acid substitutions in the E2 envelope glycoprotein." J Virol 86(11): 6084-6096.
- Hallengärd, D. et al. (2014) 'Novel attenuated Chikungunya vaccine candidates elicit protective immunity in C57BL/6 mice.', Journal of virology. American Society for Microbiology (ASM), 88(5), pp. 2858–66. doi: 10.1128/JVI.03453-13.
- Her, Z., Y. W. Kam, et al. (2009). "Chikungunya: a bending reality." Microbes Infect 11(14-15): 1165-1176.
- Hochedez, P., S. Jaureguiberry, et al. (2006). "Chikungunya infection in travelers." <u>Emerg Infect Dis</u> **12**(10): 1565-1567.
- Hoke, C. H., Jr., J. Pace-Templeton, et al. (2012). "US Military contributions to the global response to pandemic chikungunya." <u>Vaccine</u> **30**(47): 6713-6720.
- Marimoutou, C., J. Ferraro, et al. (2015). "Chikungunya infection: self-reported rheumatic morbidity and impaired quality of life persist 6 years later." <u>Clin Microbiol Infect</u> 21(7): 688-693.
- McClain, D. J., P. R. Pittman, et al. (1998). "Immunologic interference from sequential administration of live attenuated alphavirus vaccines." <u>J Infect Dis</u> **177**(3): 634-641.
- NIAID (October 26, 2016 ). "Emerging Infectious Diseases/Pathogens." https://www.niaid.nih.gov/research/emerging-infectious-diseases-pathogens.

- Pialoux, G., B. A. Gauzere, et al. (2007). "Chikungunya, an epidemic arbovirosis." <u>Lancet Infect Dis</u> **7**(5): 319-327.
- Ramsauer, K., M. Schwameis, et al. (2015). "Immunogenicity, safety, and tolerability of a recombinant measles-virus-based chikungunya vaccine: a randomised, double-blind, placebo-controlled, active-comparator, first-in-man trial." <u>Lancet Infect Dis</u> **15**(5): 519-527.
- Reisinger, Emil C. et al. 2018. "Immunogenicity, Safety, and Tolerability of the Measles-Vectored Chikungunya Virus Vaccine MV-CHIK: A Double-Blind, Randomised, Placebo-Controlled and Active-Controlled Phase 2 Trial." The Lancet 392(10165): 2718–27. http://dx.doi.org/10.1016/S0140-6736(18)32488-7.
- Reeza, G. Weaver S.C. (2019). "Chikungunya as a paradigm for emerging viral diseases: Evaluating disease impact and hurdles to vaccine development." PLoS Negl Trop Dis. 201913(1):e0006919
- Robinson, M. C. (1955). "An epidemic of virus disease in Southern Province, Tanganyika Territory, in 1952-53. I. Clinical features." <u>Trans R Soc Trop Med Hyg</u> **49**(1): 28-32.
- Schrauf, Sabrina, Roland Tschismarov, Erich Tauber, and Katrin Ramsauer. 2020. "Current Efforts in the Development of Vaccines for the Prevention of Zika and Chikungunya Virus Infections." Frontiers in Immunology 11(April): 1–20.
- Simizu, B., K. Yamamoto, et al. (1984). "Structural proteins of Chikungunya virus." <u>J Virol</u> **51**(1): 254-258.
- Simon, F., E. Javelle, et al. (2015). "French guidelines for the management of chikungunya (acute and persistent presentations). November 2014." Med Mal Infect 45(7): 243-263.
- Simon, F., E. Javelle, et al. (2015). "Chikungunya Virus Infections." N Engl J Med 373(1): 93-94.
- Simon, F., H. Savini, et al. (2008). "Chikungunya: a paradigm of emergence and globalization of vector-borne diseases." Med Clin North Am **92**(6): 1323-1343, ix.
- Suhrbier, A., M. C. Jaffar-Bandjee, et al. (2012). "Arthritogenic alphaviruses--an overview." Nat Rev Rheumatol 8(7): 420-429.
- Voss, J. E., M. C. Vaney, et al. (2010). "Glycoprotein organization of Chikungunya virus particles revealed by X-ray crystallography." Nature **468**(7324): 709-712.
- Weaver, S. C. and M. Lecuit (2015). "Chikungunya virus and the global spread of a mosquito-borne disease." N Engl J Med 372(13): 1231-1239.
- Weaver, S. C., J. E. Osorio, et al. (2012). "Chikungunya virus and prospects for a vaccine." <u>Expert Rev Vaccines</u> **11**(9): 1087-1101.